Protocol Addendum J4E-MC-FR01 (c)

A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, 52-Week Study

to Evaluate the Efficacy and Safety of LY3454738 in the Treatment of Adult Patients with

Moderate-to-Severe Atopic Dermatitis

NCT05911841

Approval Date: 06-May-2024

# **Title Page**

## **Confidential Information**

The information contained in this document is confidential and is intended for the use of clinical investigators. It is the property of Eli Lilly and Company or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of LY3454738, unless such persons are bound by a confidentiality agreement with Eli Lilly and Company or its subsidiaries.

**Note to Regulatory Authorities:** This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

**Master Protocol Title:** A Master Protocol for Randomized, Controlled, Phase 2 Clinical Trials of Multiple Interventions for the Treatment of Adults with Moderate-to-Severe Atopic Dermatitis

**Master Protocol Number:** J4E-MC-IMMB(b)

**ISA Title:** A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, 52-Week Study to Evaluate the Efficacy and Safety of LY3454738 in the Treatment of Adult Patients with Moderate-to-Severe Atopic Dermatitis

ISA Number: J4E-MC-FR01 ISA Amendment Number: c

Compound: LY3454738

**ISA Brief Title:** A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, 52-Week Study to Evaluate the Efficacy and Safety of LY3454738 in the Treatment of Adult Patients with Moderate-to-Severe Atopic Dermatitis

**Study Phase: 2** 

Sponsor Name: Eli Lilly and Company

Legal Registered Address: Eli Lilly and Company, Indianapolis, Indiana, USA 46285

**Regulatory Agency Identifier Numbers:** 

IND: 163615

EU trial number: 2022-502888-38-00

Approval Date: ISA Amendment (c) Electronically Signed and Approved by Lilly on date

provided below.

**Document ID:** VV-CLIN-150737

Medical monitor name and contact information will be provided separately.

# **Protocol Amendment Summary of Changes Table**

| DOCUMENT HISTORY | |
|-------------------|-------------|
| Document | Date |
| Amendment (b) | 12-Sep-2023 |
| Amendment (a) | 13-Mar-2023 |
| Original Protocol | 09-Dec-2022 |

## Amendment [c]

This amendment is considered to be substantial.

The amendment is considered to be substantial because it is likely to have a significant impact on the

- safety or rights of the study participants
- reliability and robustness of the data generated in the clinical study, and
- conduct or management of the trial.

#### **Overall Rationale for the Amendment**

The main purpose of this amendment is to

- collect more data in **CCI** patients, and
- revise the interim plan.

| Section # and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 1.1. Synopsis (Objectives, Endpoints, and Estimands) 3. Objectives, Endpoints, and Estimands | The secondary endpoint for efficacy is CCI CCI Studied for that objective. Added additional secondary objective and endpoint for CCI CCI participants as "Proportion of CCI | To collect more information about CCI CCI CCI |

| Section # and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 9.3.3. Secondary<br>Endpoints/Estimands<br>Analysis | Added the analyses methods CCI CCI EASI-75 at Week 16. | |
| 1.1. Synopsis (Study Population) 4.1. Overall Design 9.5. Sample Size Determination | (Text with strikethrough is replaced by text in bold) The text is updated to include the change in study population which is an addition of 60 CCI CCI | To collect more information about CCI in atopic dermatitis. |
| 9.2. Analyses Sets | Added CCI CCI population in Maintenance Analysis Set. | |
| 9.5. Sample Size Determination | With the updated planned sample size, the text is updated | |

| Section # and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| | as "an EASI-75 response at Week 16 of CCI CCI CCI 98% power for pairwise comparisons with placebo." | |
| 1.1. Synopsis (Study Population) | (Text with strikethrough is replaced by text in bold) | To allow to over enroll if needed. |
| 9.5. Sample Size Determination | "Up to CCI<br>CCI<br>CCI | |
| 1.1. Synopsis<br>(Number of<br>Participants)<br>9.5. Sample Size<br>Determination | (Text with strikethrough is deleted) "Up to approximately 260 participants will be randomized to study intervention." | |
| 1.3. Schedule of Activities | A new row for estimated glomerular filtration rate (eGFR) is added which will be determined at Week 16, Week 40, and ED Visits. | To monitor kidney function throughout the study. |
| 4.1. Overall Design | The randomization text is updated and the text below is added to include the changes in the CCI CCI CCI | |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| | CCI | |
| 4.1. Overall Design<br>9.5. Sample Size<br>Determination | The table is revised to include the updated planned sample CCI | |



# CONFIDENTIAL

# **Table of Contents**

| l. | Protocol Summary | |
|---|---|---|
| 1.1. | Synopsis | 11 |
| 1.3. | Schedule of Activities (SoA) | 18 |
| 2. | Introduction | |
| 2.1. | Study Rationale | |
| 2.2.<br>2.3. | Background | |
| 2.3.1. | Benefit/Risk Assessment | |
| 2.3.1. | Benefit Assessment | |
| 2.3.2. | Overall Benefit Risk Conclusion | |
| 3. | Objectives, Endpoints, and Estimands | |
| 3.1. | Estimands | |
| 4. | Study Design | 38 |
| 4.1. | Overall Design | |
| 4.2. | Scientific Rationale for Study Design | 40 |
| 4.2.1. | Patient Input into Design | 41 |
| 4.3. | Justification for Dose | 41 |
| 4.4. | End of Study Definition | 42 |
| <b>5.</b> | Study Population | 43 |
| 5.1. | ISA-Specific Inclusion Criteria | 43 |
| 5.2. | ISA-Specific Exclusion Criteria | 43 |
| 5.3. | Lifestyle Considerations | |
| 5.4. | Screen Failures | 46 |
| 5.5. | Criteria for Temporarily Delaying Randomization of a | 1.6 |
| | Participant | |
| 6. | Study Intervention(s) and Concomitant Therapy | 47 |
| 6.1. | Study Intervention(s) Administered | |
| 6.1.1. | Medical Devices | |
| 6.1.2. | Background Therapy | |
| 6.2. | Preparation, Handling, Storage, and Accountability | |
| 6.3.<br>6.4. | Assignment to Study Intervention | |
| 6.5. | Blinding Study Intervention Compliance | |
| 6.6. | Dose Modification | |
| 6.7. | Continued Access to Study Intervention after the End of the | |
| 0.7. | Study | 49 |
| 6.8. | Treatment of Overdose | |
| 6.9. | Prior and Concomitant Therapy | 50 |
| 6.9.1. | Rescue Medication | |
| 6.9.2. | Permitted Concomitant Therapy | 51 |
| 6.9.3. | Prohibited Concomitant Therapy | 51 |

| <b>7.</b> | Discontinuation of Study Intervention and Participant | |
|---|---|---|
| | Discontinuation/Withdrawal | 53 |
| 7.1. | Discontinuation of Study Intervention | 53 |
| 7.1.1. | Temporary Discontinuation of Study Intervention | 53 |
| 7.1.2. | Permanent Discontinuation of Study Intervention | |
| 7.2. | Participant Discontinuation/Withdrawal from the Study | 53 |
| 7.3. | Lost to Follow up | 53 |
| 8. | Study Assessments and Procedures | 54 |
| 8.1. | Efficacy Assessments | |
| 8.2. | Safety Assessments | 55 |
| 8.2.1. | Vital Signs | 55 |
| 8.2.2. | Physical Examinations | 55 |
| 8.2.3. | Skin Assessment with Fitzpatrick Scale of Skin Phototypes | 55 |
| 8.2.4. | Electrocardiograms | 55 |
| 8.2.5. | Chest Imaging | 56 |
| 8.2.6. | Clinical Safety Laboratory Tests | 56 |
| 8.2.7. | Pregnancy Testing. | 57 |
| 8.2.8. | Tuberculosis Testing and Monitoring | 57 |
| 8.2.9. | Hepatitis B Testing and Monitoring. | 57 |
| 8.2.10. | Hepatitis C Testing | 57 |
| 8.2.11. | Hepatic Safety Testing and Monitoring | |
| 8.2.12. | Suicidal Ideation and Behavior Risk Screening and Monitoring | 57 |
| 8.3. | Adverse Events, Serious Adverse Events, and Product | |
| | Complaints | |
| 8.3.1. | Adverse Events of Special Interest | 58 |
| CCI | | |
| 8.5. | Pharmacodynamics | |
| 8.6. | Genetics | 60 |
| 8.8. | Immunogenicity Assessments. | 60 |
| 8.9. | Medical Resource Utilization and Health Economics | |
| 9. | Statistical Considerations | |
| 9.1.<br>9.1.1. | Statistical Hypotheses | |
| - | Multiplicity Adjustment | |
| 9.2. | Analyses Sets | |
| 9.3.<br>9.3.1. | General Considerations | |
| 9.3.1. | Primary Endpoints/Estimands Analysis | |
| 9.3.2. | Filmary Endpoints/Estimands Anarysis | 03 |
| CU | | |
| 9.3.5. | Safety Analyses | 66 |
| 9.3.6. | Other Analyses | 66 |
| CCI | | |
| 9.5. | Sample Size Determination | 68 |
| 10. | Attachments to the ISA | 69 |

| 10.1. | Attachment 1: Clinical Laboratory Tests | 69 |
|---------|--------------------------------------------------------------|----|
| 10.1.1. | Clinical Laboratory Tests Performed During This ISA | 70 |
| CCI | | |
| 10.2. | Attachment 2: Contraceptive and Barrier Guidance | 75 |
| 10.2.1. | Definitions | |
| 10.2.2. | Contraception Guidance | 75 |
| 10.2.3. | Pregnancy Testing Guidance | |
| 10.3. | Attachment 3: ISA-Specific Stopping Rules | 77 |
| 10.4. | Attachment 4: Country-specific Requirements | 78 |
| 10.5. | Attachment 5: Provisions for Changes in Study Conduct During | |
| | Exceptional Circumstances. | 79 |
| CC | | |
| 10.8. | Attachment 8: Abbreviations and Definitions | 86 |
| 10.9. | Attachment 9: ISA Amendment History | 90 |
| 11. | References | 93 |

## 1. Protocol Summary

## 1.1. Synopsis

**ISA Title:** A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, 52-Week Study to Evaluate the Efficacy and Safety of LY3454738 in the Treatment of Adult Patients with Moderate-to-Severe Atopic Dermatitis

**ISA Brief Title:** A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, 52-Week Study to Evaluate the Efficacy and Safety of LY3454738 in the Treatment of Adult Patients with Moderate-to-Severe Atopic Dermatitis

## **Regulatory Agency Identifier Number(s):**

IND: 163615

EU trial number: 2022-502888-38-00

#### **Rationale:**

LY3454738 is a humanized IgG4-variant monoclonal antibody (mAb) that binds to and agonizes the human inhibitory checkpoint CD200R. CD200R is expressed on many cell types involved in the pathogenesis of atopic dermatitis (AD).

with an agonist mAb is a potential therapeutic strategy for AD and other inflammatory disorders. This study will evaluate the safety and efficacy of LY3454738 in adults with moderate-to-severe AD.

Study J4E-MC-FR01 (FR01) is a Phase 2 study to evaluate the efficacy and describe the safety of LY3454738 in adult patients with moderate-to-severe AD. Results of this study will be used to guide the dose selection for future studies and to further characterize the benefit/risk profile of LY3454738. Study FR01 is an ISA of the master IMMB protocol.

## Objectives, Endpoints, and Estimands:



## **Overall Design**

This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group, outpatient dose-ranging study to evaluate the efficacy and describe the safety of LY3454738 as compared to placebo during a 16-week induction period in adult participants with moderate-to-severe AD using these induction dosing regimens given CCI

- LY3454738 CCl mg CCl
   LY3454738 CCl mg CCl
   LY3454738 CCl mg CCl and
- placebo **CCI**

The blinded week maintenance treatment period begins CCI Participants having at least an CCI response at Week 16 will receive a maintenance dosing regimen, also CCI as listed here.

| Week 16 responders who were originally | |
|---|---|
| randomized to this induction regimen | Will receive this maintenance regimen: |
| LY3454738 CCI mg CCI | by rerandomization in column ratio: |
| <b>—</b> - | LY3454738 CO mg CC or |
| | placebo |
| LY3454738 CCI mg CCI | LY3454738 CC mg CC |
| LY3454738 <sup>66</sup> mg <b>CC</b> | LY3454738 CCI mg CCI |
| placebo | placebo CCI |

The maintenance period includes an "escape arm" for participants whose EASI response suggests the need for a higher dose. The escape therapy is LY3454738 CC mg CCI A participant will receive this escape therapy under the conditions listed here.

| Begin LY3454738 CC as escape therapy | if the participant |
|---|---|
| At Week 16 | has not achieved an <b>CC</b> response at Week 16. |
| At Weeks CCI | has not achieved an CCI response at Weeks |
| | CCI |

A participant receiving escape therapy will continue receiving escape therapy through the last dosing visit of the study (Week unless the participant is discontinued from study intervention.

Topical rescue medication is permitted (not required) in the induction period from Week 8 until Week 16 for participants who do not achieve an CCl response. In the maintenance period, use of topical rescue medication is permitted (not required) from Week until the end of the study for participants who do not achieve an CCl response. Participants who receive at least 2 doses of escape therapy at 2 consecutive visits will be permanently discontinued from study intervention if they fail to achieve an CCl response.

This study design includes investigator and participant blinding (masking). An internal assessment committee (IAC) will exist for the purpose of reviewing safety data in an unblinded fashion.

In summary, Study FR01 includes 4 study periods over a total study duration of approximately weeks:

- Screening: from CCl days prior to randomization at Week 0 (Study Day 1)
- Treatment Period Induction: from randomization at Week 0 (Study Day 1) through assessments at Week 16
- Treatment Period Maintenance: from dose administration at Week 16 CCI and
- Posttreatment Follow-Up: 2 visits, the last visit being CCI after randomization CCI

#### **Brief Summary:**

Activating CD200R with an agonist monoclonal antibody is a potential therapeutic strategy for atopic dermatitis and other inflammatory disorders.

The purpose of this study is to measure improvement in atopic dermatitis signs and symptoms after treatment with various dosing regimens of CCI administered LY3454738 compared to placebo in adult participants with moderate-to-severe atopic dermatitis.

• The LY3454738 dosing regimens to be compared to placebo in this study are these:

| <b>Induction Period</b> | Maintenance Period |
|-------------------------|----------------------|
| LY3454738 CC mg CC | LY3454738 CC mg CC |
| LY3454738 CCI mg CCI | LY3454738 CC mg CC |
| LY3454738 cc mg CCl | LY3454738 CCI mg CCI |

- The total study duration for a participant is approximately **CCl** weeks, inclusive of the screening period, treatment periods, and posttreatment follow-up period.
- Treatment is administered from Study Day 1 (randomization visit [Week 0]) through the last dose given at Week in the maintenance period.
- After Study Day 1, the visit frequency is approximately CCI for the first 16 weeks, specifically, at Weeks CCI Note: Not every visit includes administration of a treatment dose. Posttreatment follow-up visits occur at Week CCI CCI

#### **Study Population:**

The study population of Study FR01 includes adult male or female participants from 18 to 70 years of age, inclusive, who have a diagnosis of atopic dermatitis which is moderate to severe as measured by

- Eczema Area and Severity Index (EASI) score CG
- $vIGA-AD^{\mathbb{R}}$  score  $\geq 3$ , and
- $\geq$ 10% of body surface area (BSA) involvement (per EASI BSA).

Based on the entry criteria of the master IMMB protocol, participants in Study FR01 must also be candidates for systemic therapy and have a history of inadequate response to, or intolerance to, topical medications.

Participants will be excluded from Study FR01 if they

- have used certain atopic dermatitis treatments during a specified time period ("washout period") before the first dose of study intervention
- are unstable with respect to use of chronic treatments to improve sleep, and
- are unsuitable for study participation due to medical history or a current serious health condition.



#### **Number of Participants:**

Approximately 260 participants will be randomized to study intervention.

#### **Intervention Groups and Duration:**

The study includes 4 periods over a total study duration of approximately weeks. These are the treatment groups from randomization at Week 0 and until Week 16:

- LY3454738 CC mg CCI
   LY3454738 CC mg CCI
   LY3454738 CC mg CCI
   placebo CCI
- Participants having at least an CCI response at Week 16 will receive a maintenance dosing regimen, as listed here.

| Week 16 responders who were originally | |
|---|---|
| randomized to this induction regimen | Will receive this maintenance regimen: |
| LY3454738 CCI mg CCI | by rerandomization in column ratio: |
| <del>_</del> | LY3454738 CO mg CC or |
| | placebo |
| LY3454738 CC mg CC | LY3454738 CCI mg CCI |
| LY3454738 co mg CCI | LY3454738 COI mg CCI |
| placebo | placebo CC |

Maintenance dosing continues up to and including Week

Participants will receive LY3454738 CCI as "escape therapy" if they

- have not achieved an CCI response at Week 16, or
- have not achieved an CCI response at Weeks CCI

Once started, escape therapy continues through the last dosing visit of the maintenance period.

Topical rescue medication is permitted from Week 8 until Week 16 for participants who do not achieve an CCl response; topical rescue medication started during the induction period should be stopped at, or before, Week 16. Likewise, during the maintenance period, topical rescue medication is permitted from Week until the end of the study for participants who do not achieve an CCl response.

#### **Ethical Considerations of Benefit/Risk:**

CCI

Based on available clinical and nonclinical data, there are no anticipated risks that would require safety monitoring in this study beyond what is typical for clinical studies involving humanized mAbs. The administration of therapeutic monoclonal antibodies to humans can be associated with CCI

Efficacy results from a Phase 1 study support the hypothesis that LY3454738 has the potential to treat atopic dermatitis. Taking into account the measures taken to minimize risk to participants in this study, and in the context of the cumulative knowledge of LY3454738, the benefit/risk balance for participants in this Phase 2 study is assessed to be acceptable.

Data Monitoring Committee: Yes (Internal Assessment Committee).



# 1.3. Schedule of Activities (SoA)

| Table 1. Activities for screen | | | | | | - | s of St | udy J4 | E-M | C-FR0 | 1. | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| For activities at unscheduled v | visit or early o | liscont | inuatio | n visit, | see Ta | ıble 2. | | | | | | |
| Week | $\mathbb{CC}$ | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| | CCI | | | | | | | | | | | Minimum interval between Visit 401 of the |
| Visit interval tolerance | | | ±1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | master IMMB protocol and Study Day 1: |
| (window) in days | Study Day | | -1 | | | | ±3 | | | | | Participants doing CCI 15 days |
| | 1 | | | | | | | | | | | All other participants: 8 days |
| CRF visit number | V0 | | C | | | | | | | | | |
| Consent and demographics | | | | | | | | | | | | |
| | | | | | | | | | | | | Signed, documented consent for ISA FR01 |
| Informed consent | (V) | | | | | | | | | | | must be obtained before any ISA-specific tests |
| Informed consent | (X) | | | | | | | | | | | or procedures are performed. Relevant ICF may |
| | | | | | | | | | | | | be signed up to 90 days before Study Day 1. |
| | | | | | | | | | | | | Inclusion and exclusion criteria of both the |
| Inclusion and exclusion | | | | | | | | | | | | master IMMB protocol and this ISA must be |
| criteria: confirmation of | | X | | | | | | | | | | confirmed before participant is randomized to a |
| eligibility | | A | | | | | | | | | | study intervention and receives a first dose. See |
| Cligionity | | | | | | | | | | | | Section 5 of this ISA. See also Section 5 of the |
| | | | | | | | | | | | | master IMMB protocol. |
| Prespecified medical history | | X | | | | | | | | | | Eye Disease History form. |
| Concomitant medications | | X | X | X | X | X | X | X | X | X | X | Rescue medication and background emollients |
| | | 11 | 11 | | 11 | 11 | <b>4 1</b> | - 1 | 11 | 11 | 1 | are documented as concomitant medications. |
| | | | | | | | | | | | | AE collection begins when the master protocol |
| Adverse events (AEs) | | X | X | X | X | X | X | X | X | X | X | ICF is signed. CCl events will be |
| Transfer events (Tibb) | | 1 | 1 | 1 | 1 | '` | <b>4 L</b> | 1. | 1 | 1 | 1 | solicited at each visit. For AESIs, additional |
| | | | | | | | | | | | | data are collected. See Section 8.3.1. |
| Physical evaluation | | | | | | | | | | | | |
| Weight | | X | | | | | | | | | X | |

| For activities at unscheduled v | | liscont | inuatio | n visit, | see Ta | ble 2. | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | CCL | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance<br>(window) in days | Study Day | _ | ±1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | Minimum interval between Visit 401 of the master IMMB protocol and Study Day 1: • Participants doing CCI 15 days • All other participants: 8 days |
| CRF visit number | V0 | | C( | | | | | | | | | |
| Symptom-directed physical assessment | | X | | | | | | | | | X | Perform as shown here and as needed based on participant status and standard of care. May be performed by qualified personnel per local regulations. Assess for TB risk factors, and for signs and symptoms of active TB, including an assessment of peripheral lymph nodes. See Sections 8.2.2 and 8.2.8 of the master IMMB protocol. |
| Vital signs | | X | X | X | X | X | X | X | X | Х | X | Includes pulse rate, blood pressure, respiratory rate, and body temperature. Measured after the participant has been sitting at least 5 minutes. See Section 8.2.1 of the master IMMB protocol. |
| ECG 12-lead (single) (local) | | | | | | | | | | | X | A local ECG will be collected according to instructions in Section 8.2.4 of the master IMMB protocol. |
| Patient-reported outcomes (electronic) | | | | | | | | | | | | Complete prior to any clinician-administered assessments. |
| Dermatology Life Quality<br>Index (DLQI) | | X | | | X | | X | | X | | X | |
| Patient-Oriented Eczema<br>Measure (POEM) | | X | | | X | | X | | X | | X | |
| SCORing Atopic Dermatitis (subjective) (SCORAD) | | X | X | X | X | | X | | X | | X | |

| Table 1. Activities for screen | _ | | | | | - | s of St | udy J | E-M | C-FR0 | 1. | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| For activities at unscheduled | | liscont | inuatio | n visit, | see Ta | ıble 2. | | | | | | |
| Week | -CCI | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| X7* *4 * 4 1 1 | CCI | | | | | | | | | | | Minimum interval between Visit 401 of the |
| Visit interval tolerance (window) in days | Ct. de Des | _ | ±1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | master IMMB protocol and Study Day 1: • Participants doing CC 15 days |
| (window) in days | Study Day | | | | | | | | | | | All other participants: 8 days |
| CRF visit number | V0 | ı | C | | | | | | | | | |
| Atopic Dermatitis Control | | Ι | | | | | | | | | | |
| Tool (ADCT) | | X | | | X | | X | | X | | X | |
| Hospital Anxiety | | X | | | X | | X | | X | | X | |
| Depression Scale (HADS) | | Λ | | | Λ | | Λ | | Λ | | Λ | |
| Patient-reported outcomes | | | | | | | | | | | | |
| (paper) | | | | | | | | | | | | |
| Asthma Control | | X | | | | | | | | | X | |
| Questionnaire-5 (ACQ-5) | | | | | | | | | | | | |
| Clinician-administered | | | | | | | | | | | | |
| assessments (electronic) | | X | 37 | 37 | 37 | | 37 | | 37 | | 37 | |
| vIGA-AD | | X | X | X | X | | X | | X | | X | |
| Eczema Area and Severity<br>Index (EASI) | | X | X | X | X | | X | | X | | X | |
| SCORing Atopic Dermatitis (objective) (SCORAD) | | X | X | X | X | | X | | X | | X | |
| Fitzpatrick Scale of Skin<br>Phototypes | | X | | | | | | | | | | |
| Clinician-administered | | | | | | | | | | | | |
| assessments (paper) | | | | | | | | | | | | |
| Columbia-Suicide Severity | | | | | | | | | | | | AE collection should occur prior to collection |
| Rating Scale (C-SSRS) | | X | | | X | | X | | X | | X | of the C-SSRS. Adapted for the assessment of |
| Since Last Assessed | | | | | | | | | | | | ideation and behavior categories only. |

| Table 1. Activities for screen | ning/haseline | and ir | nductio | n tres | tment | neriod | s of St | ndv .I4 | 1F.M | C-FR0 | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| For activities at unscheduled v | _ | | | | | - | S 01 5t | uuy 57 | *15-1VI | C-PRO | 1. | |
| Week | CCI | | | , | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance<br>(window) in days | Study Day | _ | ±1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | Minimum interval between Visit 401 of the master IMMB protocol and Study Day 1: • Participants doing CC 15 days • All other participants: 8 days |
| CRF visit number | V0 | | C( | | | | | | | | | |
| Participant diary (electronic) | | | | | | | | | | | | |
| Diary dispense | | | | | | | | | | | | Diary is dispensed during Visit 401 of the master IMMB protocol. Diary contains the following assessments: CCI Atopic Dermatitis Sleep Scale, and Skin Pain Numeric Rating Scale. |
| Diary review | | X | X | X | X | X | X | X | X | X | X | Diary contains the following assessments: CCI Atopic Dermatitis Sleep Scale (ADSS), and Skin Pain Numeric Rating Scale (Skin Pain NRS). |

| Table 1. Activities for screen | ning/baseline | and in | ductio | n trea | tment | period | s of St | udy J4 | 4E-M | C-FR0 | 1. | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| For activities at unscheduled | _ | | | | | - | | | | | | |
| Week | | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance<br>(window) in days | Study Day | _ | ±1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | Minimum interval between Visit 401 of the master IMMB protocol and Study Day 1: • Participants doing CC 15 days • All other participants: 8 days |
| CRF visit number | V0 | | C | | | | | | | | | |
| Diary return | | (X) | | | | | | | | | | Collect diary only from participants who are not eligible for randomization (screen failed). |
| Participant education | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | |
| Diary education | (X) | | | | | | | | | X | | Education is provided at Visit 401 of the master IMMB protocol and as shown for this ISA. Additional education can be provided as needed at any time. |
| Laboratory tests and sample collections | | | | | | | | | | | | Collect before dosing unless otherwise specified. |
| Hematology | | X | | | X | | X | | X | | X | |
| Clinical chemistry | | X | | | X | | X | | X | | X | |
| Urine or serum pregnancy test (local) | | X | | | X | | X | | X | | X | For WOCBP, a pregnancy test must be performed, with the result available within 24 hours prior to dosing (see Section 8.2.7 of this ISA and Section 8.2.7 of the master IMMB protocol). Additional pregnancy tests should be performed at any time if a menstrual period is missed, or there is clinical suspicion of pregnancy, or as required by local law or regulation. |

| Table 1. Activities for screen | | | | | | | s of St | udy J | E-M | C-FR | )1. | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| For activities at unscheduled v | visit or early o | lisconti | inuatio | n visit, | see Ta | ble 2. | | | | | | |
| Week | $\mathbb{CCI}$ | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance<br>(window) in days | Study Day | _ | ±1 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | Minimum interval between Visit 401 of the master IMMB protocol and Study Day 1: • Participants doing CC 15 days • All other participants: 8 days |
| CRF visit number | V0 | | C | | | | | | | | | |
| Immunogenicity (ADA) samples | | X | X | | X | | | | X | | X | On dosing visits, collect samples before dosing. Collect additional samples at specified times relative to onset of COllect events (see Section 8.3.1.1 and Attachment 1, Section 10.1.2). |
| Stored samples | | | | | | | | | | | | |
| Genetics sample | | X | | | | | | | | | | Sample can be obtained at or after Study Day 1 |
| CC | | | | | | | | | | | | |
| Randomization and | | | | | | | | | | | | |
| dosing-related activities | | | | | | | | | | | | |
| Register visit with IWRS | | X | X | X | X | X | X | X | X | X | X | |
| Randomization to study intervention via IWRS | | X | | | | | | | | | | |
| Rerandomization via IWRS | | | | | | | | | | | X | |
| Dispense study intervention via IWRS | | X | | X | X | X | X | X | X | X | X | No dose is given at Week 1. The dose dispensed at Week 16 is the first dose of the maintenance period. |
| Administer study intervention | | X | | X | X | X | X | X | X | X | X | No dose is given at Week 1. |

Week

Study day

Weight

assessment

8.2.8 of the master IMMB

protocol.

| Table 2. Activities for mainte | | - | | | - | - | | | tinuatio | on visit, and <b>u</b> | unscheduled | visit (Study J4E-MC-FR01). |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Note: The posttreatment follow Week | y-up vis | sits are | required | d for al | l random | ized par | ticipant | S. | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance (window) in days | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | 1 | ±7 | ±7 | |
| CRF visit number | CCI | | | | | | | ED | _ | V808 | V812 | |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | Includes pulse rate, blood pressure, respiratory rate, and body temperature. Measured after the participant has been sitting at least 5 minutes. See Section 8.2.1 of the master IMMB protocol. |
| ECG 12-lead (single) (local) | | | X | | | | X | X | | | X | A local ECG will be collected according to instructions in Section 8.2.4 of the master IMMB protocol. |
| Patient-reported outcomes (electronic) | | | | | | | | | | | | Complete prior to any clinician-administered assessments. |
| Dermatology Life Quality<br>Index (DLQI) | X | X | X | X | X | X | X | X | | X | X | |
| Patient-Oriented Eczema<br>Measure (POEM) | X | X | X | X | X | X | X | X | | X | X | |
| SCORing Atopic Dermatitis (subjective) (SCORAD) | X | X | X | X | X | X | X | X | X | X | X | |
| Atopic Dermatitis Control<br>Tool (ADCT) | X | X | X | X | X | X | X | X | | X | X | |
| Hospital Anxiety Depression<br>Scale (HADS) | X | X | X | X | X | X | X | X | | X | X | |

| | | _ | | | _ | - | | | tinuatio | on visit, and | unscheduled v | visit (Study J4E-MC-FR01). |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Note: The posttreatment follow | v-up vi | sits are | require | d for al | l random | ized par | ticipant | s. | | | | |
| Week | | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance<br>(window) in days | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | _ | _ | ±7 | ±7 | |
| CRF visit number | CCI | | | | | | | ED | | V808 | V812 | |
| Patient-reported outcomes (paper) | | | | | | | | | | | | |
| Asthma Control<br>Questionnaire-5 (ACQ-5) | | | | | | X | | | | | X | |
| Clinician-administered assessments (electronic) | | | | | | | | | | | | |
| vIGA-AD | X | X | X | X | X | X | X | X | X | X | X | |
| Eczema Area and Severity<br>Index (EASI) | X | X | X | X | X | X | X | X | X | X | X | |
| SCORing Atopic Dermatitis (objective) (SCORAD) | X | X | X | X | X | X | X | X | X | X | X | |
| Fitzpatrick Scale of Skin<br>Phototypes | | | | | | | | | | | | Not performed in these study periods. |
| Clinician-administered assessments (paper) | | | | | | | | | | | | |
| Columbia-Suicide Severity<br>Rating Scale (C-SSRS) Since<br>Last Assessed | X | X | X | X | X | X | X | X | X | X | X | AE collection should occur prior to collection of the C-SSRS. Adapted for the assessment of ideation and behavior categories only. |
| Participant diary (electronic) | | | | | | | | | | | | |

| Table 2. Activities for maint | enance | and po | osttreat | ment f | ollow-up | period | s, early | discon | tinuatio | on visit, and t | unscheduled | visit (Study J4E-MC-FR01). |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Note: The posttreatment follow | v-up vi | sits are | require | d for al | l random | ized par | ticipant | s. | | | | |
| Week | | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance (window) in days | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | _ | ±7 | ±7 | |
| CRF visit number | CCI | | | | | | | ED | _ | V808 | V812 | |
| Laboratory tests and sample collections | | | | | | | | | | | | Collect before dosing unless otherwise specified. |
| Hematology | | | X | | | X | | X | | X | X | |
| Clinical chemistry | | | X | | | X | | X | | X | X | |
| Urine or serum pregnancy test (local) | X | X | X | X | X | X | X | X | | X | X | For WOCBP, a pregnancy test must be performed, with the result available within 24 hours prior to dosing (see Section 8.2.7 of this ISA and Section 8.2.7 of the master IMMB protocol). Additional pregnancy tests should be performed at any time if a menstrual period is missed, or there is clinical suspicion of pregnancy, or as required by local law or regulation. |
| Urinalysis | | | | | | X | | X | | | X | |
| Estimated glomerular filtration rate (eGFR) | | | | | | X | | X | | | | Calculated using Chronic<br>Kidney Disease Epidemiology<br>Collaboration (CKD-EPI)<br>Creatinine Equation (2021). |

| Visit interval tolerance (window) in days ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±0 W812 W812 Only for participants who are anti-HBc positive at Visit 401 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 W812 <t< th=""><th>Visit interval tolerance (window) in days ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±3 ±0 — ±7 ±7 ±7 ±7 ED — V808 V812 Only for participants who are anti-HBc positive at Visit 401 (see Section 8.2.9 of the master)</th><th>Week</th><th></th><th></th><th></th><th></th><th></th><th></th><th></th><th></th><th></th><th></th><th></th><th>Comment</th></t<> | Visit interval tolerance (window) in days ±3 ±0 — ±7 ±7 ±7 ±7 ED — V808 V812 Only for participants who are anti-HBc positive at Visit 401 (see Section 8.2.9 of the master) | Week | | | | | | | | | | | | Comment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (window) in days CRF visit number ED — V808 V812 Only for participants who are anti-HBc positive at Visit 401 (see Section 8.2.9 of the master) | (window) in days ±3 - - ±7 ±7 CRF visit number ED — V808 V812 Hepatitis B virus (HBV) X X X X Only for participants who are anti-HBc positive at Visit 401 (see Section 8.2.9 of the master) | • • | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Hepatitis B virus (HBV) X X X X Only for participants who are anti-HBc positive at Visit 401 (see Section 8.2.9 of the master) | Hepatitis B virus (HBV) X X X X Only for participants who are anti-HBc positive at Visit 401 (see Section 8.2.9 of the master) | | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | _ | _ | ±7 | ±7 | |
| Hepatitis B virus (HBV) NA X X X Anti-HBc positive at Visit 401 (see Section 8.2.9 of the master | Hepatitis B virus (HBV) DNA X X X Anti-HBc positive at Visit 401 (see Section 8.2.9 of the master) | CRF visit number | CCI | | | | | | | ED | _ | V808 | V812 | |
| | | | | X | | | X | | | X | | | X | anti-HBc positive at Visit 401 (see Section 8.2.9 of the maste |
| | | | | | _ | | | | | | | | | |

| Table 2. Activities for mainte | | | | | | | | | tinuatio | on visit, and | unscheduled | visit (Study J4E-MC-FR01). |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Note: The posttreatment follow | v-up vi | sits are | required | d for al | l random | ized par | ticipant | S. | | | | |
| Week | | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance<br>(window) in days | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | _ | _ | ±7 | ±7 | |
| CRF visit number | CCI | | | | | | | ED | _ | V808 | V812 | |
| Immunogenicity (ADA) samples | | | X | | | X | | X | | | X | On dosing visits, collect samples before dosing. Collect additional samples at specified times relative to onset of events (see Section 8.3.1.1 and Attachment 1, Section 10.1.2). |
| Stored samples | | | | | | | | | | | | , |
| Genetics sample | | | | | | | | | | | | Sample can be obtained at or after Study Day 1. |
| Randomization and dosing-related activities | | | | | | | | | | | | |
| Register visit with IWRS | X | X | X | X | X | X | X | X | | X | X | |
| Dispense study intervention via IWRS | X | X | X | X | X | X | | | | | | The last dose is given at Week 40. |

| Table 2. Activities for mainte | nance | and po | sttreati | ment f | ollow-up | period | s, early | discon | tinuatio | n visit, and | unscheduled v | isit (Study J4E-MC-FR01). |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Note: The posttreatment follow | -up vi | sits are | required | d for al | l random | ized par | ticipants | S. | | | | _ |
| Week | | | | | | | | | | | | Comment |
| Study day | | | | | | | | | | | | Study Day 1 is day of first dose. |
| Visit interval tolerance | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | | ±7 | ±7 | |
| (window) in days | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | | ±/ | ±/ | |
| CRF visit number | CCI | | | | | | | ED | _ | V808 | V812 | |
| Administer study | X | X | X | X | X | X | | | | | | The last dose is given at |
| intervention | Λ | Λ | Λ | Λ | Λ | Λ | | | | | | Week |

Abbreviations: ADA = anti-drug antibodies; AESI = adverse event of special interest; anti-HBc = hepatitis B core antibody; CRF = case report form; DNA = deoxyribonucleic acid; ECG = electrocardiogram; ED = early discontinuation visit; ICF = informed consent form; ISA = intervention-specific appendix; IWRS = interactive web-response system; TB = tuberculosis; UV = unscheduled visit; V = case report form visit; WOCBP = women of childbearing potential.

# 2. Introduction

# 2.1. Study Rationale

LY3454738 is a humanized IgG4-variant mAb that binds to and agonizes the human inhibitory checkpoint CD200R. CD200R is expressed on many cell types involved in the pathogenesis of AD. CCI

Activating CD200R with an agonist mAb is a potential therapeutic strategy for AD and other inflammatory disorders. This study will evaluate the safety

## 2.2. Background

Immune checkpoint regulators such as CD200R are critical modulators of the immune system, allowing the initiation of a productive immune response and preventing the onset of autoimmunity by negatively regulating the response once the pathogen is eliminated.

and efficacy of LY3454738 in adults with moderate-to-severe AD.

CD200R is expressed on multiple cell types. Specifically, CD200R is expressed on the surface of myeloid cells (mast cells, basophils, macrophages, and dendritic cells), and on T cells, B cells, neutrophils, microglia, and retina (Broderick et al. 2002; Wright et al. 2003). The CD200R ligand, CD200, is expressed on the surface of a variety of cell types, including vascular endothelial cells, fibroblasts, T and B cell subsets, and neurons (Wright et al. 2003).

The pathogenesis of AD involves dysregulation of adaptive and innate immune responses. Skin-resident cells such as dendritic cells, mast cells, keratinocytes, macrophages, and innate lymphoid cells contribute to the inflammation of skin in AD. Likewise, T cells, plasmacytoid dendritic cells, monocytes, and granulocytes also contribute to AD pathology (Egawa and Weniger 2015). CD200R is expressed on many of these cell types. Hence, activating CD200R with an agonist mAb such as LY3454738 is a potential strategy for the treatment of AD.

#### 2.3. Benefit/Risk Assessment

#### 2.3.1. Risk Assessment

## Risks associated with LY3454738

No dose-limiting safety issues have been identified in clinical studies of participants receiving single or repeat doses of LY3454738. In a Phase 1 study comparing LY3454738 versus placebo in AD (Study FRCC),

Based on these data and on other available clinical and nonclinical data, there are no anticipated risks that would require safety monitoring in this study beyond what is typical for clinical studies involving humanized mAbs.

The administration of therapeutic mAbs to humans can be associated with **CC** 

## CCI

## Risks and discomforts associated with study procedures

Participants will use additive-free emollients during the study but will refrain from other topical AD treatments, with the exception of rescue medication as described in Section 6.9.1. Participants accustomed to using TCS and other topical treatments may experience increased discomfort due to itching during the study.

#### Risk mitigations

The study entry criteria of the master IMMB protocol and of this ISA exclude potential participants who may be at greater risk of developing infections, CCI or malignancies. Participants who may be at greater risk for adverse effects related to TCS withdrawal (Hajar et al. 2015) are also excluded.

To reduce the burden of untreated AD symptoms, qualifying participants are permitted to receive rescue medication during certain study periods (Sections 4.1 and 6.9.1).

All participants will have appropriate predose safety assessments, including symptom-directed physical assessments, clinical safety laboratory tests, suicidality/self-harm evaluations, vital signs, and evaluation of reported AEs, during the treatment period. The design includes posttreatment follow-up visits at which safety assessments are also conducted.



#### 2.3.2. Benefit Assessment



Participants may benefit by receiving personal health information from the physical examinations and from other routine safety assessments performed in this study.

#### 2.3.3. Overall Benefit Risk Conclusion

Taking into account the measures taken to minimize risk to participants in this study, and in the context of the cumulative knowledge of LY3454738, the benefit/risk balance for participants in this Phase 2 study is assessed to be acceptable.

More detailed information about the known and expected benefits and risks and reasonably expected adverse events of LY3454738 may be found in the IB.

# 3. Objectives, Endpoints, and Estimands

This table lists objectives and endpoints for the evaluation of LY3454738 versus placebo.






### 3.1. Estimands

The primary clinical question of interest is: in the target patient population, what is the difference between each dosing regimen of LY3454738 and placebo in achieving a successful response at Week 16 without use of any prohibited or rescue medication for AD or early permanent discontinuation?

The estimand is described by the following attributes:

- Population: participants with moderate-to-severe AD.
- Endpoint: The primary endpoint and all secondary efficacy endpoints, that is,
   EASI-75 CCI
- How to account for ICEs:

- Population-level summary:
  - For binary endpoints CCI
    CCI
    the population-level summary will be the unconditional difference in response rate at Week 16 between each dosing regimen of LY3454738 and placebo.
  - o For continuous endpoints (percent change from baseline in EASI CCI mean difference at Week 16 between each dosing regimen and placebo.
- Rationale for estimand: The composite estimand is the standard from prior AD studies CCI
   CCI
   From the perspective of ICEs:
  - o If a participant used any prohibited or rescue medication for AD, the participant was not receiving sufficient benefits from study intervention.
  - o If a participant early discontinued study intervention, the participant experienced a burden of study intervention that outweighed its benefits.

### ISA: J4E-MC-FR01(c)

# 4. Study Design

# 4.1. Overall Design

This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group, outpatient dose-ranging study to evaluate the efficacy and describe the safety of multiple LY3454738 induction and maintenance dosing regimens in adult participants with moderate-to-severe AD. The study population includes participants, all with diagnosed AD which is

moderate to severe as measured by EASI score  $\geq$ 16, vIGA-AD score  $\geq$ 3, and  $\geq$ 10% of BSA involvement at randomization.

### **Study periods**

A schematic of the design of this ISA is presented CCl Assessments, sample collections, and study drug administrations occur at the visits shown in the SoA (Section 1.3).

### Screening period and randomization to treatment within this ISA (Visit 0)

Screening for this ISA can begin up to days before Study Day 1 (day of first dose). Informed consent for participation in this ISA must be obtained before any ISA-specific tests or procedures are performed. Screening activities for this ISA are listed in the SoA (Section 1.3) in the columns for CRF Visit 0 (V0).

Before a participant is randomized to a study intervention, the participant's eligibility according to the study entry criteria of both the master IMMB protocol (Section 5) and this FR01 ISA (Section 5) must be confirmed.



#### Blinded induction period

Randomized participants will begin the double-blind, placebo-controlled, 16-week induction period when the initial dose is administered on Study Day 1.

Topical rescue medication is permitted from Week 8 until Week 16 for participants who do not achieve an CCI response, as described in Section 6.9.1. Topical rescue medication started during the induction period should be stopped at, or before, Week 16.

### Blinded maintenance period

The blinded —-week maintenance treatment period begins with the dose administered at Week 16. Participants having at least an CCI response at Week 16 will receive a maintenance dosing regimen, as listed here.

| Week 16 responders who were originally | |
|---|---|
| randomized to this induction regimen | Will receive this maintenance regimen: |
| LY3454738 CCI mg CCI | by rerandomization in <sup>CCI</sup> ratio: LY3454738 <sup>CCI</sup> mg CCI or |
| | placebo |
| LY3454738 CCI mg CCI | LY3454738 CCI mg CCI |
| LY3454738 <sup>cc.</sup> mg <b>CC</b> | LY3454738 CCI mg CCI |
| placebo | Placebo CCI |

The maintenance period includes an "escape arm" for participants whose EASI response suggests the need for a higher dose. The escape therapy is LY3454738 [CC] mg [CC]. A participant will receive this escape therapy under the conditions listed here.

| Begin LY3454738 CC mg CC as escape therapy | if the participant |
|---|---|
| At Week 16 | has not achieved an CCI response at Week 16. |
| At Weeks CC | has not achieved an CC response at Weeks CC |
| | CCI |

A participant receiving escape therapy will continue receiving escape therapy through the last dosing visit of the study (Week unless the participant is discontinued from study intervention.

Topical rescue medication in the maintenance period is permitted from Week until the end of the study for participants who do not achieve an celebrate response, as described in Section 6.9.1.

### Posttreatment follow-up period

All participants are expected to have 2 follow-up visits after the last dosing visit, as listed here.

| Condition | First follow-up visit | Second follow-up visit |
|---|---|---|
| If the participant did not discontinue | occurs approximately 8 wk after | occurs approximately 12 wk after |
| study intervention early | last dosing visit | last dosing visit |
| If the participant <b>did</b> discontinue study | occurs after ED and with an | occurs after ED and with an |
| intervention early | approximately 8-week interval | approximately 12-week interval |
| | between the last dose and this | between the last dose and this visit |
| | visit | |

#### **Blinding**

This study design includes investigator and participant blinding (masking) (Section 6.4). Blinding of the participant's original induction and maintenance treatments will continue until all participants have completed their last posttreatment follow-up visit or have discontinued the study. All blinded assessments and sample collections should be completed before a dose is administered at the dosing visits.



#### **Internal assessment committee**

During the study, an IAC will review the safety data in an unblinded fashion, as described in the master IMMB protocol, Appendix 1, Section 10.1.5.

# 4.2. Scientific Rationale for Study Design

### EASI-75 as the primary endpoint measure

The EASI and SCORAD are both regarded as acceptable instruments to measure the clinical signs of AD (Schmitt et al. 2013). Study FR01 uses a 75% reduction relative to the baseline EASI score (EASI-75) as the primary measure of efficacy. The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD (Hanifin et al. 2001).

### Duration of treatment period and posttreatment follow-up

The duration of the induction period (16 weeks) and the primary endpoint at Week 16 is based on previous clinical trials of systemic therapies in AD (Simpson et al. 2016). The remaining duration of the study is intended to allow exploratory assessments of various LY3454738

maintenance dosing regimens. To reduce participant burden, topical rescue medication is permitted under certain circumstances (Section 6.9.1).

The posttreatment follow-up period allows for continued monitoring of safety and maintenance of response after the last dose. The duration of this period is considered sufficient to wash out LY3454738 based on the half-life of the CCI mg dose, CCI

### Appropriateness of study population

The study inclusion criteria will enable enrollment of patients who are representative of the general population with moderate-to-severe AD. The EASI score  $\geq$ 16, IGA score  $\geq$ 3, and  $\geq$ 10% of BSA involvement at baseline have been used as inclusion criteria in other studies of AD (Simpson et al. 2016).

#### Choice of placebo control, number of treatment groups, and escape arm

A double-blind, placebo-controlled design limits bias for the participant assessments and investigator assessments and enables a clearer interpretation of the effects of the active study intervention.

The multiple dosing regimens enable an evaluation of safety and efficacy across several doses and frequencies, thereby providing information to guide the selection of dosing regimens for future studies.

The maintenance "escape arm" for nonresponders gives participants an opportunity to remain in the study and receive potential benefit from a higher dose.

### 4.2.1. Patient Input into Design

Not applicable.

#### 4.3. Justification for Dose

The LY3454738 dose range of mg to mg to is based on clinical safety data from the Phase I Study FRCC, CCI The chosen dose levels and regimens are anticipated to provide an exposure range that is pharmacologically active and cover a range of clinical response.





In the maintenance period, **CCI** regimens of LY3454738 and placebo are included to determine whether less frequent dosing can maintain the response attained with **CCI** induction dosing regimens.

# 4.4. End of Study Definition

A participant is considered to have completed this FR01 ISA if the participant has completed all periods of the study, including the last scheduled procedure shown in the SoA of this ISA (Section 1.3).

The end of this ISA is defined as the date of the last scheduled procedure of the last participant in Study FR01 globally.

# 5. Study Population

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

All screening evaluations, including those specified in the master IMMB protocol, must be completed and reviewed to confirm that each potential participant meets all eligibility criteria (that is, both master protocol and ISA-specific criteria) before the participant is randomized and receives the first dose of study intervention in this ISA.

The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

### 5.1. ISA-Specific Inclusion Criteria

Participants are eligible to be included in this ISA only if all of the following criteria apply.

#### **Informed consent**

- [1000] Are capable of giving, and have given, signed informed consent, which includes consent to compliance with the requirements and restrictions listed in the ICF(s) and in this ISA, including compliance with the use of contraceptives as specified in this ISA (see Attachment 2, Section 10.2.2).
- [1001] Are considering and capable of undergoing the study procedures applicable to the participant's study site.

### Participant characteristics

[1002] Are from 18 to 70 years of age (inclusive) at the time of signing the ICF(s).

### **Disease-specific characteristics**

[1003] Have moderate-to-severe AD, defined as meeting all of the following criteria, at the first dosing visit:

```
[1003a] EASI score \geq16
[1003b] vIGA-AD score \geq3, and
[1003c] \geq10% of BSA involvement (per EASI BSA).
```

[1004] Have applied at least 1 emollient every day for at least 2 weeks before the day of the first dose of study intervention in this ISA and agree to daily use of at least 1 emollient continuously throughout the study.

# 5.2. ISA-Specific Exclusion Criteria

Participants are excluded from this ISA if any of the following criteria apply.

[1005] Have, in the screening period (Visit 0), any of the skin conditions, infections, or medical conditions listed in Section 5.2 of the master IMMB protocol.

# Previous or current therapies

[1006] Have received any of the following therapies during the specified time period ("washout") or are anticipated to need any of these therapies during the study:

| Criterion | Therapy | Time period ("washout") before the first dose of study intervention <sup>a</sup> | Note |
|---|---|---|---|
| C | | | |
| [1006b] | Corticosteroids that are • parenteral (administered via intra-articular, intramuscular, or IV route), or • rectally administered (enemas or suppositories) | 6 weeks | Intranasal, inhaled, or ophthalmic (ocular) steroids are allowed at any time. |
| [1006c] | Oral systemic corticosteroids | 4 weeks | |
| [1006e] | Other systemic therapy used to treat AD or symptoms of AD, whether approved/marketed or off-label use | 4 weeks | |
| [1006f] | Any investigational CC | 4 weeks or 5 half-lives (whichever is longer) | |
| [1006g] | Phototherapy, including • therapeutic phototherapy (psoralen plus ultraviolet A, ultraviolet B) • excimer laser, or • tanning beds | 4 weeks | |
| [1006h] | Topical immune modulators, including TCIs (for example, tacrolimus, pimecrolimus), and JAK inhibitors (for example, ruxolitinib, delgocitinib) | 2 weeks | |
| [1006i] | PDE4 inhibitors (for example, crisaborole) | 2 weeks | |
| [1006j] | Bleach bath | 2 weeks | |
| [1006k] | TCS | 2 weeks | |

- a The washout period in this table includes the day of the first dose of study intervention.
- [1007] Have received any live vaccine (that is, live attenuated) within less than 4 weeks before the day of the first dose of study intervention in this ISA, or intend to receive a live vaccine during the study, or within 14 weeks (about 5 half-lives) after receiving the last dose of study intervention.

Note: The following are not considered live vaccines: RNA vaccines, vaccines with inactive viral elements, and/or nonreplicating viral vector vaccines. Nonlive SARS-CoV-2 vaccines authorized by local regulatory bodies are allowed during or after the study.

- [1008] Have received a BCG vaccination or treatment within less than 4 weeks before the day of the first dose of study intervention in this ISA, or intend to receive BCG vaccination or treatment during the study, or within 14 weeks after receiving the last dose of study intervention.
- [1009] Are unstable with respect to use of chronic treatments to improve sleep:
  - [1009a] Have started or restarted using a prescription sleep medication during the 2 weeks before the day of the first dose of study intervention in this ISA
  - [1009b] Have changed the dose of a prescription sleep medication during the 2 weeks before the day of the first dose of study intervention in this ISA, or
  - [1009c] Are likely to need to start or change the dose of prescription sleep medication during this ISA, in the opinion of the investigator.

Note: Individuals on a stable dose of prescription sleep medication at screening may be eligible to be enrolled if other study entry criteria are met, but such individuals should remain on the stable dose throughout the study unless, in the investigator's opinion, the dose should be changed or stopped to address a safety concern (Section 6.9.2).

### Other previous or current medical conditions

- [1010] Have 1 or more of the following conditions suggesting a possibly greater risk of clinically significant CCI reactions:
  - [1010a] known CC LY3454738, related compounds, or any components of the formulation, or
  - [1010b] history of CCI reactions that in the opinion of the investigator may predispose the participant to a clinically significant to LY3454738 or to any components of the formulation.

### Previous or concurrent clinical trial participation

[1011] Have received LY3454738 in any other clinical study.

#### Other

[1012] Are unable or unwilling to make themselves available for the required number of study visits or are unwilling to follow study restrictions and procedures, including restrictions on the use of concomitant therapies for AD, such as TCS.

### **5.3.** Lifestyle Considerations

Participants should be instructed not to donate blood or blood products for 18 weeks after their last dose of study intervention.

Participants must agree to the contraception criteria detailed in Attachment 2, Section 10.2.2, of this ISA, and they must agree not to breastfeed at any time during the study.

#### 5.4. Screen Failures

Individuals who do not meet the criteria for participation in this ISA (screen failure at the ISA level) cannot be rescreened for this same ISA (FR01) using the same participant number.

See the master IMMB protocol for additional information.

# 5.5. Criteria for Temporarily Delaying Randomization of a Participant

Not applicable. See the master IMMB protocol.

# 6. Study Intervention(s) and Concomitant Therapy

Study intervention is defined as any medicinal product or medical device intended to be administered to or used by a study participant according to the study protocol.

### 6.1. Study Intervention(s) Administered

This study involves placebo and dose levels of LY3454738 administered with CCl shown in this table.

| Intervention Name | LY3454738 | Placebo CC |
|---|---|---|
| Nominal Dose Levels | CCI mg | Not applicable |
| | ccl mg | |
| | CCI mg | |
| | mg mg | |
| Frequency of Administration | CCI<br>CCI | and as needed to maintain the blind |
| Route of Administration | CCI | CCI |
| Authorized as defined by EU | Not authorized | Authorized and not used according to |
| Clinical Trial Regulation | | authorization |

Abbreviations: EU = European Union; CCl

Background therapy will be used as shown in this table.

| Intervention Name | <b>Background therapy:</b> emollient without additives such as |
|---|---|
| | antiprurities or antiseptics, as described in Section 6.1.2 of the |
| | master IMMB protocol |
| Dose Levels | Per local approved label, if applicable |
| Frequency of Administration | Daily or per local approved label, if applicable |
| Route of Administration | Topical |
| Authorized as defined by EU Clinical | Not authorized <sup>a</sup> |
| Trial Regulation | |

Abbreviation: EU = European Union.

LY3454738 will be supplied for clinical trial use as a CCI
The drug product vials will be supplied in cartons, with the appropriate quantity specific to the planned dispensing schedule.

### Preparing the study interventions for dosing

An unblinded pharmacist or other unblinded qualified individual will prepare the study interventions CCI (see Section 6.4).



a This medicinal product is not authorized in accordance with Directive 2001/83/EC and Regulation (EC) No 726/2004 of the European Parliament and of the Council. However, emollients are authorized according to EU Regulation 1223/2009 and are being used according to their authorization.



### Monitoring of participants after dosing

All participants should be monitored for 30 minutes or longer after dosing, according to investigator practice or local standard of care. Sites must have resuscitation equipment, emergency drugs, and appropriately trained staff available during the completion of all required postdosing activities.

### Supply and labeling of study interventions

See the master IMMB protocol.

#### **6.1.1.** Medical Devices

Not applicable to this ISA.

### 6.1.2. Background Therapy

See the master IMMB protocol.

# 6.2. Preparation, Handling, Storage, and Accountability

See the master IMMB protocol.

# **6.3.** Assignment to Study Intervention

Assignment to treatment groups within this ISA will be determined by a computer-generated random sequence using an IWRS. The randomization ratios are described in Section 4.1.

The randomization will be stratified based on the following factors:



- baseline disease severity: baseline vIGA-AD 3 versus baseline vIGA-AD 4, and
- sex assigned at birth: male or female.

# 6.4. Blinding

This is a double-blind study. Participants, investigators, and all individuals involved in the treatment or clinical evaluation of the participants will remain blinded to each participant's original induction and maintenance treatments until all participants have completed their last posttreatment follow-up visit or have discontinued the study.

The switching of an individual participant to the escape arm is not blinded. The investigator will be aware of each participant's EASI response and of the fact that participants meeting certain EASI criteria (specified in Section 4.1) will be switched to LY3454738 [CCI] mg [CCI] as escape therapy. The participant's original induction and maintenance treatments will nevertheless remain blinded until all participants have completed their last posttreatment follow-up visit or have discontinued the study.

### Use of an unblinded pharmacist

To maintain the blind, persons otherwise uninvolved in the study, for example, unblinded pharmacists or other unblinded qualified individuals, will prepare the study interventions When LY3454738 is prepared for dosing according to the detailed instructions provided by the sponsor, it will not be possible to distinguish LY3454738 from placebo.

Blinded study personnel will administer the study intervention to the participants.

### **Emergency unblinding**

See the master IMMB protocol.

### 6.5. Study Intervention Compliance

The date and time of each dose administered will be recorded in the source documents and will be recorded in the CRF. The dose of study intervention and study participant identification will be confirmed prior to the time of dosing. Deviations from the prescribed dosage regimen are identifiable via the CRF.

#### 6.6. Dose Modification

The dosing regimens used in this study are described in Sections 4.1 and 6.1. No modifications to the specified regimens (dose or frequency) are permitted, except for reasons of immediate participant safety.

# 6.7. Continued Access to Study Intervention after the End of the Study

Continued access to the study interventions of this ISA will not be provided to participants after they have finished participating in this ISA.

### **6.8.** Treatment of Overdose

An overdose of LY3454738 is considered to be any dose greater than the highest dose of LY3454738 planned for use in this study.

In the event of an actual or suspected overdose, the investigator should

- contact the medical monitor immediately
- evaluate the participant to determine, in consultation with the medical monitor, whether study intervention should be interrupted or whether the dose should be reduced, and

• closely monitor the participant for any AE/SAE and laboratory abnormalities as medically appropriate for at least 14 weeks. Hematology, chemistry, vital signs, and oxygen saturation should be monitored and supportive care should be provided as necessary (see the IB for LY3454738).

## 6.9. Prior and Concomitant Therapy

See the master IMMB protocol for general instructions about recording any vaccine, therapy, or medication that the participant receives during the study.

#### **6.9.1.** Rescue Medication

### Rescue medication during induction period

If a participant meets this criterion during this time period, the decision to implement rescue medication is per the investigator's judgment and is not a protocol requirement. Rescue medication started during this period must be stopped at the Week 16 visit.

### Rescue medication during maintenance and posttreatment follow-up periods

Use of rescue medication is permitted **starting at Week** and until the end of the study for participants who **do not achieve an** response. If a participant meets this criterion during this time period, the decision to implement rescue medication is per the investigator's judgment and is not a protocol requirement.

#### Medications for use as rescue

This table lists the allowed rescue medications.

| Allow | ed as rescue medication <sup>a</sup> | Alternative or limitation |
|---|---|---|
| • | triamcinolone 0.1% cream | If these are not available, an alternate, equivalent potency TCS |
| • | hydrocortisone 2.5% ointment, or | cream or ointment can be used. |
| • | both | |
| • | TCIs | If these are prescribed, their use should be limited to problem |
| • | crisaborole, or | areas only, for example, face, neck, skin folds, and genital areas. |
| • | both | |

a Rescue medications should be used according to their local product labeling.

Abbreviations: TCI = topical calcineurin inhibitor; TCS = topical corticosteroid.

### Additional medications and considerations for use as rescue

This table describes additional medications and considerations for use as rescue.

| If a participant | then |
|---|---|
| does not improve sufficiently after using | a higher potency TCS may be used. |
| the specified rescue medication for 7 days | |
| reaches "clear" to "almost clear" skin | the medium- and/or high-potency TCS and TCI should be |
| after rescue with medium- and/or | stopped, and a low-potency TCS, for example, hydrocortisone |
| high-potency TCS and TCI | 2.5% ointment, should be used once daily for an additional |
| | 7 days, and then stopped. |

| If a participant | then |
|---|---|
| has lesions return after stopping rescue | retreat with TCS with or without TCIs and/or crisaborole as |
| | before, at the discretion of the investigator. |

#### Time of administration of rescue medication

Investigators should make every attempt to conduct efficacy and safety assessments immediately before administering any rescue medication. An unscheduled visit can be used for this purpose if necessary. This is to allow adequate assessment of skin dryness at the visit.

#### **Documentation of rescue medication**

Rescue medication must be recorded as stated in Section 6.9 of the master IMMB protocol.

### Discontinuation due to inadequate control with rescue medication

Participants receiving rescue medication will continue to receive the assigned study interventions. A participant should be discontinued from study intervention and proceed to the posttreatment follow-up period if, in the investigator's judgment, there is inadequate response to rescue medication, as specified in Section 7.1.2.

### 6.9.2. Permitted Concomitant Therapy

### Permitted concomitant therapies for AD

Concomitant therapies for AD during the study are permitted only as described here:

- Daily use of emollients is required as background therapy, as described in Section 6.1 and Section 6.1.2 of the master IMMB protocol.
- Rescue medication (for example, triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment; TCIs and/or crisaborole; medium- and/or high-potency TCS and TCI) is permitted but not required, as described in Section 6.9.1.
- Use of topical and oral nonsedating antihistamines is permitted.

### Permitted concomitant therapies for other conditions

Concomitant therapies for conditions other than AD are generally allowed unless described as prohibited in Section 6.9.3. Here is guidance for some of the permitted concomitant therapies:

- Intranasal or inhaled steroids: Use of intranasal or inhaled steroids is allowed at any time for participants with such conditions as asthma and allergic rhinitis.
- Prescription sleep medications: Individuals on a stable dose of prescription sleep medication at screening should remain on this stable dose throughout the study unless, in the investigator's opinion, the dose should be changed or stopped to address a safety concern.

### **6.9.3.** Prohibited Concomitant Therapy

Medications and treatments prohibited before randomization to a study intervention are listed in the exclusion criteria of this ISA (Section 5.2).

This table lists therapies prohibited throughout the study, that is, from randomization until the last posttreatment follow-up visit of this ISA.

**Prohibited Concomitant Therapy** Note Systemic corticosteroids, including, but not limited to, Note: Intranasal or inhaled or ophthalmic (ocular) oral or parenteral corticosteroids (intra-articular, steroid use is allowed at any time (Section 6.9.2). intramuscular, IV, or rectally administered) Phototherapy, including therapeutic phototherapy (psoralen plus ultraviolet A, ultraviolet B), excimer laser, and tanning beds Any investigational therapy except the study interventions used in this ISA CBD products and any of the following substances if medically prescribed for the treatment of symptoms of AD or other conditions: marijuana, marijuana extract, and THCs-containing products Bleach baths Allergen immunotherapy • The following are not considered live vaccines: RNA vaccines, vaccines with inactive viral elements, and/or nonreplicating viral vector Nonlive SARS-CoV-2 vaccines authorized by local Live vaccines or BCG vaccination regulatory bodies are allowed during or after the • Live vaccines and BCG vaccination are prohibited both during the study and within 14 weeks after the last dose of study intervention.

Abbreviations: AD = atopic dermatitis; BCG = Bacillus Calmette-Guerin; CBD = cannabidiol; IV = intravenous; JAK = Janus kinase; RNA = ribonucleic acid; TCS = topical corticosteroid; THC = tetrahydrocannabinol.

# 7. Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal

### 7.1. Discontinuation of Study Intervention

See the master IMMB protocol.

### 7.1.1. Temporary Discontinuation of Study Intervention

See the master IMMB protocol.

#### 7.1.1.1. Elevated Liver Test Results

See the master IMMB protocol.

### 7.1.2. Permanent Discontinuation of Study Intervention

Possible reasons for permanent discontinuation of study drug include, but are not limited to, the reasons listed here as well as reasons listed in Section 7.1.2 of the master IMMB protocol.

- Inadequate response to rescue medication in participants who have been receiving rescue medication: at the **second** of **2** consecutive visits, the investigator determines that rescue medication is inadequate to control the participant's AD symptoms and the participant needs treatment with an AD therapy which is prohibited by the protocol. In such cases, the participant is to be discontinued from the study drug before starting the protocol-prohibited AD therapy.
- Nonresponse in participants who are receiving escape therapy: Participant receiving at least 2 doses of escape therapy at 2 consecutive visits fails to achieve an CCI response.

# 7.2. Participant Discontinuation/Withdrawal from the Study

See the master IMMB protocol.

### 7.3. Lost to Follow up

See the master IMMB protocol.

### ISA: J4E-MC-FR01(c)

### 8. Study Assessments and Procedures

Study procedures and their timing are summarized in the SoAs of the master IMMB protocol and this ISA. Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct. Since key efficacy and patient-reported outcomes data may be collected via an electronic tablet and/or diary, adherence to the data collection modality specified in the SoA is also essential and is required for study conduct.

Unless otherwise specified in the SoA of this ISA, all blinded assessments and sample collections should be completed before a dose is administered at the dosing visits.

# 8.1. Efficacy Assessments

Efficacy-related assessments occur at visits specified in the SoA of this ISA (Section 1.3).

See Appendix 6, Section 10.6, of the master IMMB protocol for descriptions of these assessments:

- EASI
- vIGA-AD
- SCORAD
- POEM
- DLQI

ADCT



- ADSS
- Skin Pain NRS

This ISA also includes the ACQ-5 and HADS, which are described here.

### Asthma Control Questionnaire-5 (ACQ-5)

The ACQ-5 is a participant-reported, 5-item questionnaire that assesses the following domains:

- awoken at night by symptoms
- limitation of normal daily activities
- morning symptoms
- shortness of breath (dyspnea), and
- wheezing.

The 5 questions are scored on a 7-point Likert scale with a recall period of 1 week. The scores range from 0 to 6 (higher score = lower asthma control). The total ACQ-5 score is the mean score of all questions; a lower score represents better asthma control. The ACQ-5 has been shown to reliably measure asthma control and distinguish participants with well-controlled asthma (score  $\leq$ 0.75 points) from those with uncontrolled asthma (score  $\geq$ 1.5 points) (Juniper et al. 1999; Juniper et al. 2006).

### **Hospital Anxiety Depression Scale (HADS)**

The HADS is a validated, participant-reported instrument that assesses both anxiety and depression for the previous week. Fourteen items are rated on a 4-point scale from 0 to 3 (Zigmond and Snaith 1983; White et al. 1999). Higher numbers indicate greater dysfunction (Zigmond and Snaith 1983; Herrmann 1997; Snaith 2003).

This table describes the scoring.

| HADS Subscale | Number of <b>Questions</b> | Rating Score for<br>Each Question | Score | <b>Total Score Range</b> |
|---|---|---|---|---|
| Anxiety | 7 | 0-3 | Sum of odd items | 0-21 |
| Depression | 7 | 0-3 | Sum of the even items | 0-21 |

Total scores of each subscale greater than or equal to 8 are interpreted as potential cases.

Total scores of each subscale greater than or equal to 11 are interpreted as clinically significant symptoms (Zigmond and Snaith 1983).

# 8.2. Safety Assessments

### Visits and order of safety assessments

Safety assessments occur at visits specified in the SoA (Section 1.3) of this ISA, in addition to the screening safety assessments specified in the SoA for the master IMMB protocol.

See the master IMMB protocol for

- the preferred order of completing multiple safety assessments at the same visit (IMMB Section 8)
- general provisions for safety monitoring during the study (IMMB Section 8.2), and
- safety data collection and reporting requirements (IMMB Section 8.3).

### 8.2.1. Vital Signs

See the master IMMB protocol.

#### 8.2.2. Physical Examinations

See the master IMMB protocol for a description of

- TB assessment
- complete physical examination, and
- symptom-directed physical assessments.

Height and weight will be measured and recorded as specified in the SoA of this ISA.

### 8.2.3. Skin Assessment with Fitzpatrick Scale of Skin Phototypes

See the master IMMB protocol.

### 8.2.4. Electrocardiograms

For each participant, 12-lead ECGs will be collected as specified in the IMMB SoA (Section 1.3) and the SoA of this ISA.

See the master IMMB protocol for a description of the

- timing of collection of ECGs
- interpretation of collected ECGs
- actions to be taken after a clinically significant finding on ECGs, and
- documentation of review of ECGs.

### 8.2.5. Chest Imaging

See the master IMMB protocol.

#### 8.2.6. Clinical Safety Laboratory Tests

In this ISA, Attachment 1 (Section 10.1) and the SoA (Section 1.3) provide a list of clinical laboratory tests to be performed during this ISA. See the master IMMB protocol for clinical laboratory tests performed at Visit 401.

All protocol-required laboratory assessments, as defined in this ISA and as defined in the master IMMB protocol, must be conducted in accordance with the SoA, standard collection requirements, and the laboratory manual.

### Reviewing and recording test results

See the master IMMB protocol for instructions about reviewing and recording clinical laboratory test results.

### Repeat testing after a clinically significant abnormal finding

All laboratory tests with values considered clinically significantly abnormal during participation in the study, or within 14 weeks after the last dose of study intervention, should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the investigator or medical monitor. If such values do not return to normal/baseline within a period of time judged reasonable by the investigator, the etiology should be identified and the sponsor notified.

#### **Fasting visits**

Fasting is not required before any clinical trial visits in this study.

# Laboratory tests after CC event

See Attachment 1, Section 10.1.2, of this ISA for clinical laboratory samples to be collected after event.

### Allowance for additional laboratory testing

Additional clinical laboratory tests may be performed at any time during the study as deemed necessary by the investigator or as required by local regulations.

### 8.2.7. Pregnancy Testing

Pregnancy testing is to be performed for WOCBP at the visits specified in the SoA (Section 1.3). If the specified visit includes administration of study intervention, the pregnancy test must be "negative" within 24 hours before the study intervention is administered.

See Section 8.2.7 of the master IMMB protocol for additional information.

### 8.2.7.1. Optional FSH Testing

See the master IMMB protocol.

### 8.2.8. Tuberculosis Testing and Monitoring

See the master IMMB protocol.

### 8.2.9. Hepatitis B Testing and Monitoring.

See the master IMMB protocol.

### 8.2.10. Hepatitis C Testing

See the master IMMB protocol.

#### 8.2.11. Hepatic Safety Testing and Monitoring

See the master IMMB protocol for guidance about the close hepatic monitoring, comprehensive hepatic evaluation, and suggested actions and follow-up assessments.

# 8.2.11.1. Additional Hepatic Data Collection (Hepatic Safety CRF) in Study Participants Who Have Abnormal Liver Tests During the Study

See the master IMMB protocol.

#### 8.2.12. Suicidal Ideation and Behavior Risk Screening and Monitoring

#### Screening for suicidal ideation or behavior

Screening for suicidal ideation or behavior includes the C-SSRS, as specified in the SoA for the master IMMB protocol.

### Monitoring for suicidal ideation and behavior and depressive symptomatology

During the treatment and posttreatment periods of this ISA as specified in the SoA (Section 1.3), the C-SSRS (adapted for the assessment of ideation and behavior categories only) will be used to monitor for suicidal ideation and behavior. See the master IMMB protocol for a description of the C-SSRS.

#### Discontinuation of participants with signs of suicidal ideation or behavior

Participants who have signs of suicidal ideation or behavior should be considered for discontinuation of study intervention, following a risk assessment (see Section 7.1.2 of the master IMMB protocol).

# 8.3. Adverse Events, Serious Adverse Events, and Product Complaints

See the master IMMB protocol for instructions on

- timing and mechanism for collecting adverse events and product complaints
- adverse event monitoring with a systematic questionnaire, and
- collection of pregnancy information.

### **8.3.1.** Adverse Events of Special Interest

For this ISA, the AESIs include



If these AESIs are reported, sites will be prompted to collect additional data as described in the following subsections.

Nonleading (spontaneous) AE collection should occur before the collection of any solicited AE or AE follow-up questionnaires.





# 8.5. Pharmacodynamics

CCI

### 8.6. Genetics

Where local regulations and IRB/IEC allow, a whole blood sample will be collected from consenting participants, as specified in the SoA (Section 1.3) of this ISA, for pharmacogenetic analysis.

#### Additional information

See the master IMMB protocol for information about

- use of genetics samples
- confidentiality of genetics samples, and
- retention of genetics samples.



# 8.8. Immunogenicity Assessments

Predose venous blood samples will be collected to determine antibody production against the study intervention.

#### Collection visits and times

The visits and times for collecting samples for ADA testing are specified in the SoA (Section 1.3) of this ISA. The actual date and time (24-hour clock time) of each sample collection must be recorded accurately on the appropriate forms. To aid interpretation of these results, a venous blood sample will be collected at same time points to determine the serum concentrations of LY3454738. All samples for immunogenicity should be taken predose when applicable and possible.

Immunogenicity will be assessed by a validated assay designed to detect ADAs in the presence of LY3454738. Antibodies may be further characterized for their neutralizing ability.

# Samples collection for CCl event

If CCI event is suspected, additional blood samples will be obtained for ADA analyses, as described in Attachment 1, Section 10.1.2, of this ISA.

### **Additional information**

See the master IMMB protocol for additional information about retention of ADA samples.

# 8.9. Medical Resource Utilization and Health Economics

Health economics or medical resource utilization and health economics parameters will not be collected in this ISA.

### 9. Statistical Considerations

This section is a summary of the planned statistical analyses of the most important endpoints, including primary and secondary endpoints, of this ISA. The MP-SAP and ISA-SAP will include a more technical and detailed description of the statistical analyses described in this section. The ISA-SAP will be finalized prior to the first unblinding.

# 9.1. Statistical Hypotheses

The null hypotheses corresponding to the primary and secondary estimands are these: there is no difference between LY3454738 and placebo in participants with moderate-to-severe AD with respect to

• proportion of participants achieving EASI-75 at Week 16 (primary)



### 9.1.1. Multiplicity Adjustment

No adjustments for multiplicity will be performed.

# 9.2. Analyses Sets

For the purposes of analysis, the following analysis sets are defined:

| Analysis Set | Description | Populations | Analyses<br>Conducted on<br>This Analysis Set |
|---|---|---|---|
| Induction<br>Analysis Set | All randomized participants who receive at least 1 dose of study intervention. Participants | • Overall | <ul><li>vIGA-AD</li><li>EASI</li><li>SCORAD</li></ul> |
| | will be included in the analysis set according to their randomly assigned intervention. | | • PROs |
| Maintenance | All randomized participants | • Overall | • vIGA-AD |
| Analysis Set | who enter the maintenance<br>period. Participants will be<br>included in the analysis set<br>according to their randomly<br>assigned interventions at Week<br>0 and Week 16. | CCI | <ul><li>EASI</li><li>SCORAD</li><li>CCI</li><li>PROs</li></ul> |

| Analysis Set | Description | Populations | Analyses<br>Conducted on<br>This Analysis Set |
|---|---|---|---|
| Safety | All randomized participants receiving at least 1 dose of study intervention. Participants will be included in the analysis set according to the intervention they actually received. | • Overall | Safety data<br>analyses for<br>induction and/or<br>maintenance<br>period |
| Pharmaco-kinetics (PK) | All randomized participants receiving at least 1 dose of study intervention and have PK data available. | • Overall | PK data analyses<br>for induction<br>and/or<br>maintenance<br>period |

Abbreviations: EASI = Eczema Area and Severity Index; NRS = Numeric Rating Scale; PK = pharmacokinetic; PROs = patient-reported outcomes; SCORAD = SCORing Atopic Dermatitis.

Additional analysis sets will be defined in the ISA-SAP to support exploratory analyses.

# 9.3. Statistical Analyses

#### 9.3.1. General Considerations

Statistical analysis of this study will be the responsibility of the sponsor or its designee. All statistical tests, unless otherwise noted, will be 2-sided and will be performed at a significance level of 0.05. Unless indicated otherwise in the ISA-SAP, the analyses will be conducted as described in this section.

#### Changes to the data analysis methods

Any change to the data analysis methods described in this ISA will require an amendment only if the change affects a principal feature of the ISA. Any other change to the data analysis methods described in the ISA and the justification for making the change will be described in the CSR. Additional exploratory analyses of the data will be conducted as deemed appropriate. Complete details of the planned analyses will be documented in the ISA-SAP.

#### Summary of data

Continuous data will be summarized in terms of mean, standard deviation, minimum, maximum, median, and number of observations. Categorical data will be summarized as frequency counts and percentage. Comparison between each LY3454738 dosing regimen and placebo will be performed for all efficacy and patient-reported endpoint analyses during the induction period with no adjustment for multiple comparisons.

#### **Induction dose selection**

Dose selection at the end of the induction period will be based on comparisons between each regimen and placebo using dose-response modeling. Dose selection rules and specifics will be detailed in the ISA-SAP.

#### **Baseline definition**

For efficacy and PRO analyses, baseline will be defined as the last available value before the first dose of study intervention. In most cases, this value will be what is recorded at the randomization visit (Visit 0). For efficacy measures, if a participant does not take any study intervention, the last available value on or prior to randomization date will be used. Change from baseline will be calculated as the visit value of interest minus the baseline value.

For induction period safety analyses, the baseline period is defined as the time from Visit 401 to the first dose of study intervention. For the safety analyses during the maintenance period, baseline is defined as the last available value before the first dose of study intervention during the maintenance period. In most cases, this will be the measure recorded at Week 16. For the safety analyses during the posttreatment follow-up period, baseline is defined as the last nonmissing assessment on or prior to entering the posttreatment period, that is, on or prior to Week 44 or ED visit.

### Missing data

For the estimand defined in Section 3.1, missing data after accounting for ICEs is expected to be uncommon. Thus, the handling of any missing data remaining after accounting for ICEs will be specified in the ISA-SAP. Missing data imputation methods for supplementary estimands will be described in the ISA-SAP.

#### **Induction treatment comparisons**



#### **Maintenance treatment comparisons**

The efficacy of different maintenance regimens will primarily be assessed with descriptive statistics across the maintenance period. Frequencies and percentages will summarize binary outcomes, and means and standard deviations will summarize continuous outcomes. The ISA-SAP may include additional exploratory analyses for maintenance efficacy, including, but not limited to, inferential efficacy analyses and the efficacy of different maintenance regimens across differing levels of response at induction, for example, CCI EASI-75 responders at Week 16.

# 9.3.2. Primary Endpoints/Estimands Analysis

| Treatment comparisons between ea | ach LY3454738 dosing regimen and placebo in proportion of |
|---|---|
| CCI | participants achieving EASI-75 at Week 16 will be |
| conducted with CCI | at a significance level of 0.05. |
| The analysis will be conducted using | ng the induction analysis set CCI |
| CCI | where participants who have ICEs of interest prior to |
| Week 16 will be considered as non | responders. |

Treatment response rates, treatment differences versus placebo, and their corresponding 95% CIs will be provided according to study intervention to which participants are randomized at Visit 0.



ISA: J4E-MC-FR01(c)



### 9.3.5. Safety Analyses

See Section 9.3.5 of the master IMMB protocol for safety analyses, including but not limited to, AEs and SAEs.

### 9.3.6. Other Analyses

See the master IMMB protocol (Section 9.3.6) for participant disposition and characteristics, concomitant therapy, treatment compliance, PROs, subgroups, and sensitivity analyses.

### 9.3.6.1. Pharmacokinetic/Pharmacodynamic Analyses

Serum concentrations of LY3454738 will be listed by time point and dosing regimen using descriptive statistics. The PK of LY3454738 may also be characterized using graphical evaluations and mixed-effect (population PK) modeling approaches.



Data from this study may be combined with other study data, if appropriate. Details on PK and PK/PD analyses will be provided in an ISA-SAP or a separate ISA PK/PD analysis plan.

### 9.3.6.2. Immunogenicity Analyses

Upon assay validation, the frequency and percentage of participants with preexisting ADA and with TE ADA may be tabulated. TE ADAs are defined as those with a titer 2-fold (1 dilution) greater than the minimum required dilution, if no ADAs were detected at baseline (treatment-induced ADA) or those with a 4-fold (2 dilutions) increase in titer compared with baseline, if ADAs were detected at baseline (treatment-boosted ADA).

The frequency of neutralizing antibodies may also be tabulated in TE ADA-positive participants, when available.

The relationship between the presence of ADA and LY3454738 concentrations or PK parameters and PD response, including safety and efficacy, may be assessed.





# 9.5. Sample Size Determination

Approximately 260 participants will be randomized to study intervention.



With this planned sample size, an EASI-75 response at Week 16 of 52% and 12% for LY3454738 and placebo, respectively, CCl participants achieve at least 91% power for pairwise comparisons with placebo using a 2-sided chi-square test at the 0.05 significance level, with no adjustment for multiple comparisons.

### 10. Attachments to the ISA

This section provides information specific to the FR01 ISA. For supporting documentation and operational considerations applicable to all ISAs, see Section 10 of the master IMMB protocol.

### **10.1.** Attachment 1: Clinical Laboratory Tests

#### Use of central or local laboratories

Clinical laboratory tests will be performed by a central laboratory or by a local laboratory as detailed in the tables in this attachment.

In circumstances where the sponsor approves local laboratory testing in lieu of the central laboratory testing specified in the tables, the local laboratory must be qualified in accordance with applicable local regulations.

### Laboratory tests for inclusion/exclusion of potential study participants

See Section 5 of the master IMMB protocol for laboratory tests that are part of the master IMMB protocol eligibility criteria. See Section 5 of this ISA for additional laboratory testing (if any) that may be required to assess eligibility.

### Allowance for additional laboratory testing

Additional tests may be performed at any time during the study as determined necessary by the investigator or required by local regulations.

### **Investigator responsibilities**

Investigators must document their review of the laboratory safety results.

### Provision of laboratory test results

Laboratory test results that could unblind the study will not be reported to investigative sites or other blinded personnel.

# 10.1.1. Clinical Laboratory Tests Performed During This ISA

This section lists the clinical laboratory tests performed at the visits specified in the SoA (Section 1.3) of this ISA.

| | Notes |
|---|---|
| Hematology | Assayed by Lilly-designated laboratory. |
| Hemoglobin | |
| Hematocrit | |
| Erythrocyte count (red blood cells [RBC]) | |
| Mean cell volume | |
| Mean cell hemoglobin | |
| Mean cell hemoglobin concentration | |
| Absolute neutrophil count (ANC) (segmented and | |
| bands) (calculated) | |
| Leukocytes (white blood cells [WBC]) | |
| Differential | |
| Percent and absolute count of: | |
| Neutrophils, segmented | |
| Neutrophils, bands | Report if detected. |
| Lymphocytes | |
| Monocytes | |
| Eosinophils | |
| Basophils | |
| Platelets | |
| Cell morphology (RBC and WBC) | |

| | Notes |
|----------------------------------|-----------------------------------------|
| Clinical Chemistry | Assayed by Lilly-designated laboratory. |
| Sodium | |
| Potassium | |
| Chloride | |
| Bicarbonate | |
| Total bilirubin (TBL) | |
| Direct bilirubin | |
| Alkaline phosphatase (ALP) | |
| Alanine aminotransferase (ALT) | |
| Aspartate aminotransferase (AST) | |
| Gamma-glutamyl transferase (GGT) | |
| Blood urea nitrogen (BUN) | |
| Creatinine | |
| Creatine kinase (CK) | |
| Uric acid | |
| Total protein | |
| Albumin | |
| Calcium | |
| Phosphorus | |
| Glucose (random) | |

| | Notes |
|---|---|
| Hormones (females) | |
| Serum pregnancy | Performed locally. For WOCBP only. See Section 8.2.7. |
| Urine pregnancy | Performed locally. For WOCBP only. See Section 8.2.7. |
| Follicle-stimulating hormone (FSH) | Optional. Performed locally. See Section 8.2.7.1. |

| | Notes |
|---|---|
| Urinalysis | Assayed by Lilly-designated laboratory. |
| Specific gravity | |
| pН | |
| Protein | |
| Glucose | |
| Ketones | |
| Bilirubin | |
| Urobilinogen | |
| Blood | |
| Nitrite | |
| Urine leukocyte esterase | |
| Microscopic examination of sediment | Perform if abnormalities were detected on urinalysis. |
| | Notes |
|---|---|
| Hepatitis Serology | |
| Hepatitis B virus (HBV) testing: | Assayed by Lilly-designated laboratory. |
| | Performed only for participants who test positive for |
| Hepatitis B virus (HBV) DNA | anti-HBc at screening. |



| | Notes |
|---|---|
| | Assayed by Lilly-designated laboratory. |
| Pharmacokinetics (PK) Samples | Results will not be provided to the investigative sites. |
| LY3454738 concentration | |

| | Notes |
|---|---|
| | Assayed by Lilly-designated laboratory. |
| Immunogenicity Samples | Results will not be provided to the investigative sites. |
| Anti-LY3454738 antibodies | |
| anti-LY3454738 antibodies neutralization | |

| | Notes |
|---|---|
| | Assayed by Lilly-designated laboratory. |
| <b>Genetics Sample</b> | Results will not be provided to the investigative sites. |



Abbreviations: DNA = deoxyribonucleic acid; EDTA = ethylenediaminetetraacetic acid; RNA = ribonucleic acid; WOCBP = women of childbearing potential.



## 10.2. Attachment 2: Contraceptive and Barrier Guidance

#### 10.2.1. Definitions

See the master IMMB protocol.

#### 10.2.2. Contraception Guidance

#### **Females**

WOCBP who are completely abstinent as their preferred and usual lifestyle, or in a same-sex relationship as their preferred and usual lifestyle:

| Must | Must not |
|---|---|
| agree to either remain<br>abstinent or stay in a<br>same-sex relationship<br>without sexual<br>relationships with males | <ul> <li>use periodic abstinence methods</li> <li>calendar</li> <li>ovulation</li> <li>symptothermal, or</li> <li>postovulation</li> <li>declare abstinence just for the duration of a trial, or</li> <li>use the withdrawal method</li> </ul> |

WOCBP who are NOT completely abstinent as their preferred and usual lifestyle, or NOT in a same-sex relationship as their preferred and usual lifestyle, must do the following:

| Topic | Condition |
|---|---|
| Pregnancy testing | Have pregnancy testing at initial screening: See the master IMMB protocol. Have subsequent pregnancy testing as described in the SoA (Section 1.3) of this ISA. |
| Contraception | Agree to use 2 forms of effective contraception, where at least 1 form must be highly effective. |
| | Note: These forms of contraception must be used during the study and after the study for at least 18 weeks after the last dose of the study intervention. |

## **Examples of different forms of contraception:**

| Methods | Examples |
|---|---|
| Highly effective contraception (less than 1% failure rate) | <ul> <li>female sterilization</li> <li>combination oral contraceptive pill</li> <li>progestin-only contraceptive pill (mini-pill)</li> <li>implanted contraceptives</li> <li>injectable contraceptives</li> <li>contraceptive patch (only women &lt;198 pounds or 90 kg)</li> <li>total abstinence</li> <li>vasectomy (if only sexual partner)</li> <li>fallopian tube implants (if confirmed by hysterosalpingogram)</li> <li>combined contraceptive vaginal ring, or</li> <li>intrauterine devices</li> </ul> |
| Effective contraception | <ul> <li>male or female condoms with spermicide</li> <li>diaphragms with spermicide or cervical sponges</li> <li>barrier method with use of a spermicide <ul> <li>condom with spermicide</li> <li>diaphragm with spermicide, or</li> <li>female condom with spermicide</li> </ul> </li> <li>Note: Male and female condoms should not be used in combination.</li> </ul> |
| Ineffective forms of contraception whether used alone or in any combination | <ul> <li>spermicide alone</li> <li>periodic abstinence</li> <li>fertility awareness (calendar method, temperature method, cervical mucus, or symptothermal)</li> <li>withdrawal</li> <li>postcoital douche, or</li> <li>lactational amenorrhea</li> </ul> |

#### Males

No male contraception is required except in compliance with specific local government study requirements.

## 10.2.3. Pregnancy Testing Guidance

See Sections 1.3 and 8.2.7 of the master IMMB protocol, and Section 1.3 and Section 8.2.7 of this ISA.

## 10.3. Attachment 3: ISA-Specific Stopping Rules

The IAC will convene periodically but also when the accumulated safety data triggers one of the stopping rules specified in this ISA. Further enrollment in this ISA, or further dosing in this ISA, or both may be stopped, pending a decision of the IAC.

## **Stopping rules for Study FR01**

The IAC will evaluate unblinded safety data from Study FR01 if

- 5 or more participants experience TEAEs in the same system organ class
- these TEAEs are serious (meeting at least 1 criterion which defines SAEs) or are assessed by the investigator as severe, or both, and
- these TEAEs are considered related to the blinded study intervention in the opinion of the investigator.

# 10.4. Attachment 4: Country-specific Requirements

#### For sites in EU Member States

This attachment is not applicable at this time.

## For sites outside of EU Member States

Country-specific requirements, if any, will be described in a separate protocol addendum.

#### ISA: J4E-MC-FR01(c)

# 10.5. Attachment 5: Provisions for Changes in Study Conduct During Exceptional Circumstances

Appendix 12, Section 10.12, of the master IMMB protocol, which describes provisions for changes in study conducting during exception circumstances, is applicable to this ISA.

In addition, the changes described in this attachment are applicable. These are temporary measures intended to be used only during specific time periods as directed by the sponsor in partnership with the investigator.

See Appendix 12, Section 10.12, of the master IMMB protocol for these topics:

- exceptional circumstances
- implementing changes under exceptional circumstances
- considerations for making a change, and
- informed consent.

#### Changes in study conduct during exceptional circumstances

Changes in study conduct not described in Appendix 12, Section 10.12, of the master IMMB protocol or in this attachment, or not consistent with applicable local regulations, are not allowed. The following changes in study conduct will not be considered protocol deviations.

#### Remote visits

Types of remote visits for Visit 0 and thereafter

**Telemedicine:** Telephone or technology-assisted virtual visits, or both, are acceptable to complete appropriate assessments. Assessments to be completed in this manner may include, but are not limited to, concomitant medications, Aes, participant diary education and compliance check, and PROs via a tablet and/or a web-based collection system.

**Mobile health care:** Health care visits may be performed by a mobile health care provider at locations other than the study site when participants cannot travel to the site if written approval is provided by the sponsor. Procedures performed at such visits may include, but are not limited to, vital signs, concomitant medications, Aes, participant diary education and compliance check, symptom-directed physical assessments, ECGs, collection of blood and urine samples for clinical safety laboratory testing, C-SSRS Since Last Assessed, PROs via a tablet and/or a web-based collection system.

**Other alternative locations:** Procedures which could be done at an alternate location may include, but are not limited to, ECGs, biopsy sample collections, and collection of blood and urine samples for clinical safety laboratory testing.

See Appendix 12, Section 10.12, of the master IMMB protocol for additional information on data capture, safety reporting, and return to on-site visits.

#### Local laboratory testing option for Visit 0 (Week 0) and thereafter

Local laboratory testing may be conducted in lieu of central laboratory testing. However, central laboratory testing must be retained for samples listed in this table:

| At | Central laboratory testing must be retained for these samples |
|---|---|
| Week 0 (Visit 0) | All samples, unless local testing is specified in the SoA (Section 1.3) and |
| | Attachment 1, Section 10.1. |
| Week 16 | Hematology, clinical chemistry, and urinalysis. |
| All weeks/visits | CCI |

The local laboratory must be qualified in accordance with applicable local regulations.

## Study intervention and ancillary supplies (including participant diaries)

See Appendix 12, Section 10.12, of the master IMMB protocol.

In addition, if study intervention will be administered to the participant during a mobile health care visit or at an alternate location, there must be resuscitation equipment, emergency drugs, and appropriately trained staff available during the CCI and until completion of all required postdosing activities.

## Screening period guidance

See Appendix 12, Section 10.12, of the master IMMB protocol.

#### Adjustments to visit windows for Visit 0 (Week 0) and thereafter

Whenever possible and safe to do so, as determined by the investigator's discretion, study procedures should be completed within the visit windows described in the relevant SoA. To maximize the possibility that these visits can be conducted as on-site visits, the windows for visits may be adjusted, upon further guidance from the sponsor. This minimizes missing data and preserves the intended conduct of the study.

This table describes the allowed adjustments to visit windows.

| For this week or type of visit | the permitted visit type is | and the visit interval tolerance <sup>a</sup> is |
|---|---|---|
| | | 1 1 0 1 |
| Week 0 | on-site only | same as shown in the SoA |
| Weeks 1 though 14 | remote | same as shown in the SoA |
| Week 16 | combination of | on-site: EASI, vIGA-AD, SCORAD (clinical portion) |
| | on-site and remote | within 7 days before or within 7 days after the |
| | | targeted visit date (inclusive) |
| | | remote: other procedures, same tolerance as shown in |
| | _ | the SoA |
| | remote | same as shown in the SoA |
| CCI | combination of | on-site: EASI, vIGA-AD, SCORAD (clinical portion) |
| | on-site and remote | within 7 days before or within 7 days after the |
| | | targeted visit date (inclusive) |
| | | remote: other procedures, same tolerance as shown in |
| | | • |
| | | the SoA |
| Unscheduled | remote | not applicable |

| For this week or type of visit | the permitted visit type is | and the visit interval tolerance <sup>a</sup> is |
|---|---|---|
| Early discontinuation | combination of on-site and remote | on-site: EASI, vIGA-AD, SCORAD (clinical portion) within 7 days after the early discontinuation decision remote: other procedures, same tolerance as shown in the SoA |
| Posttreatment follow-up<br>8 weeks after ED or final<br>treatment period visit | remote | same as shown in the SoA |
| Posttreatment follow-up 12 weeks after ED or final treatment period visit | remote | same as shown in the SoA |

<sup>&</sup>lt;sup>a</sup> Note: For participants whose visits have extended windows, additional study intervention may need to be provided to avoid interruption and maintain overall integrity of the study.

#### **Documentation**

See Appendix 12, Section 10.12, of the master IMMB protocol.









# 10.8. Attachment 8: Abbreviations and Definitions

| Term | Definition |
|---|---|
| ACQ-5 | Asthma Control Questionnaire-5 |
| AD | atopic dermatitis |
| ADA | anti-drug antibodies |
| ADCT | Atopic Dermatitis Control Tool |
| ADSS | Atopic Dermatitis Sleep Scale |
| AE | adverse event |
| AESI | adverse event of special interest |
| CCI | |
| anti-HBc | hepatitis B core antibody |
| AxMP | auxiliary medicinal product. See further definition in the master IMMB protocol |
| BCG | Bacillus Calmette-Guerin |
| BSA | body surface area |
| CBD | cannabidiol |
| CI | confidence interval |
| CRF | case report form |
| CSR | clinical study report |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DLQI | Dermatology Life Quality Index |
| DNA | deoxyribonucleic acid |
| EASI | Eczema Area and Severity Index |
| CCI<br>EASI-75 | Participant's EASI score is reduced by at least CCI 75% CCI relative to their baseline score |
| ECG | electrocardiogram |
| ED | early discontinuation |

| EU | European Union |
|---------|---------------------------------------------------|
| HADS | Hospital Anxiety Depression Scale |
| HBV | hepatitis B virus |
| hr | hour or hours |
| IAC | Internal Assessment Committee |
| IB | investigator brochure |
| ICE | intercurrent event |
| ICF | informed consent form |
| IEC | independent ethics committee |
| IGA | Investigator's Global Assessment |
| CCI | |
| IND | Investigational New Drug application |
| IRB | institutional review board |
| ISA | intervention-specific appendix |
| ISA-SAP | statistical analysis plan for the ISA |
| CCI | |
| IWRS | interactive web-response system |
| JAK | Janus kinase |
| LS | least squares |
| mAb | monoclonal antibody |
| MAD | multiple-ascending dose |
| MCMC-MI | Markov Chain Monte Carlo – multiple imputation |
| CCI | |
| min | minute or minutes |
| MP-SAP | statistical analysis plan for the master protocol |

TCS

TE ADA

**TEAE** 

THC

US or USA

| NRS | Numeric Rating Scale |
|---|---|
| PC | product complaint |
| PD | pharmacodynamic |
| PDE4 | phosphodiesterase type 4 |
| PK | pharmacokinetic |
| POEM | Patient-Oriented Eczema Measure |
| PRO | patient-reported outcome |
| CCI | |
| RNA | ribonucleic acid |
| CCI | |
| SAD | single-ascending dose |
| SAE | serious adverse event |
| CCI | |
| SCORAD | SCORing Atopic Dermatitis |
| SCORAD-75<br>SCORAD-90 | Participant's SCORAD score is reduced by at least 75% or 90% relative to their baseline score |
| SoA | schedule of activities |
| CCI | |
| ТВ | tuberculosis |
| CCI | |
| TCI | topical calcineurin inhibitor |

topical corticosteroid

tetrahydrocannabinol

United States of America

treatment-emergent anti-drug antibodies

treatment-emergent adverse event

| CONFIDENTIAL | Master Protocol J4E-MC-IMMB(b) | ISA: J4E-MC-FR01(c) |
|--------------|--------------------------------|---------------------|
| | | ` ' |

| UV | unscheduled visit |
|---|---|
| V | case report form visit |
| WOCBP | women of childbearing potential; see further definition in the master IMMB protocol |

## 10.9. Attachment 9: ISA Amendment History

The Protocol Amendment Summary of Changes Table for the current amendment is located before the Table of Contents.

## **Amendment [a]: (13-Mar-2023)**

#### **Overall Rationale for the Amendment:**

The purpose of this amendment is to classify the ACQ-5 as a paper instrument, to add a secondary objective for safety, to clarify dosing instructions, and to obtain additional information about CCI Minor editorial corrections and formatting errors are not represented in this table.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 1.1. Synopsis | Added safety objective and | To improve alignment between objectives and title |
| | endpoints as secondary objective | and rationale for study |
| 1.3. Schedule of | In the Aes rows of Tables 1 and | To improve awareness of the need to obtain |
| Activities (SoA) | 2, added an instruction that | additional information about these events |
| | information about CCI | |
| | events will be solicited at | |
| | each visit | |
| 1.3. Schedule of | In Tables 1 and 2, listed ACQ-5 | To reflect the fact that the instrument will be |
| Activities (SoA) | as a paper patient-reported | provided to participants on paper, not |
| | outcomes instrument | electronically |
| 1.3. Schedule of | In Table 1, added a CCI | To have additional data for understanding |
| Activities (SoA) | at Week 16 | responder data at later time points |
| 3. Objectives, | Moved safety objective from | To improve alignment between objectives and title |
| Endpoints, and | exploratory to secondary, and | and rationale for study |
| Estimands | added safety endpoints | |
| 3.1. Estimands | Added the word "efficacy" in the | To align estimands text with changes made in |
| | phrase "secondary efficacy | Section 3 |
| | endpoints" | |
| 6. Study Intervention(s) | Reworded the definition of study | To improve alignment with regulatory definitions |
| and Concomitant | intervention | |
| Therapy | | |
| 6.1. Study | Corrected the instructions about | To clarify and correct the instructions to more |
| Intervention(s) | CCI | easily evaluate any <b>CCl</b> if they |
| Administered | CCI | occur |
| 8.3.1. Adverse Events | Added new text and a new | To obtain additional information about these |
| of Special Interest | subsection (Section 8.3.1.5) | comorbidities |
| | about the solicitation of | |
| | comorbid CCI events | |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 10.9. Attachment 9: | Revised statement about | To ensure internal document consistency |
| ISA Amendment | amendment history | |
| History | | |

## **Amendment [b]: (12-Sep-2023)**

This amendment is considered to be substantial.

The amendment is considered to be substantial because it is likely to have a significant impact on the primary or major secondary analyses.

#### **Overall Rationale for the Amendment:**

The purpose of this amendment is to

- change the primary estimand and associated statistical methodology
- change the verbiage regarding the primary database interim analysis and populating language for another interim analysis based on enrollment of CCI data, and
- remove the topical corticosteroid question.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 1.1. Synopsis 3.1. Estimands | Primary estimand was changed from a CCI estimand CCI CCI to a composite estimand for all intercurrent events (ICEs) of interest. The role of prohibited medications related to atopic dermatitis (AD) was clarified as an ICE of interest. | This change aligns the primary estimand and analysis CCI CCI |
| 1.1. Synopsis<br>(subsection Study<br>Population and Number of<br>Participants) | Added statement for 60 randomized participants who will CCICCI added "up to" to the number of participants subsection to read as "Up to approximately 260 participants will be randomized" | For better clarity |
| 1.3. Schedule of Activities (SoA) 8.1. Efficacy Assessments | Removed TCS question | The TCS question was removed to reduce burden to sites and participants and to avoid duplicated data collection with the concomitant medication forms. |
| 9.2. Analyses Sets | Added "at Week 0 and Week 16" in maintenance analysis set | For better clarity |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 9.3.1. General | The handling of missing data after | Missing data after accounting for ICEs |
| considerations | accounting for ICEs of interest in the | of interest are expected to be |
| 9.3.2. Primary | updated primary estimand will be | uncommon in the updated primary |
| Endpoints/Estimands | specified in the statistical analysis plan | estimand. |
| Analysis | for the ISA (ISA-SAP). | |
| | () | |
| CCI | | |
| 9.3.1. General | | |
| considerations | | |
| 9.3.1. General | | |
| considerations | | |
| 9.3.2. Primary | | |
| Endpoints/Estimands | | |
| Analysis | | |
| CCI | | |
| 9.5. Sample Size | Updated the language and added | For better clarity |
| Determination | number of participants | |
| 10.9. Attachment 9: ISA | Inserted date, rationale, and summary | To update document history |
| Amendment History | of changes from ISA amendment (a). | 7. 0 |
| 11. References | CCI | For reference |

## ISA: J4E-MC-FR01(c)

#### 11. References



Broderick C, Hoek, RM, Forrester JV, et al. Constitutive retinal CD200 expression regulates resident microglia and activation state of inflammatory cells during experimental autoimmune uveoretinitis. *Am J Pathol.* 2002;161(5):1669-1677. https://doi.org/10.1016/S0002-9440(10)64444-6

Egawa G, Weninger W. Pathogenesis of atopic dermatitis: a short review. *Cogent Biology*. 2015;1(1):1103459. https://doi.org/10.1080/23312025.2015.1103459



- Hajar T, Leshem YA, Hanifin JM, et al. A systematic review of topical corticosteroid withdrawal ("steroid addiction") in patients with atopic dermatitis and other dermatoses. *J Am Acad Dermatol*. 2015; 72(3): 541-549.e2. https://doi.org/10.1016/j.jaad.2014.11.024
- Hanifin JM, Thurston M, Omoto M, et al. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. *Exp Dermatol*. 2001;10(1):11-18. https://doi.org/10.1034/j.1600-0625.2001.100102.x
- Herrmann C. International experiences with the Hospital Anxiety and Depression Scale a review of validation data and clinical results. *J Psychosom Res* 1997;42(1):17-41. https://doi.org/10.1016/S0022-3999(96)00216-4
- Juniper EF, O'Byrne PM, Guyatt GH, et al. Development and validation of a questionnaire to measure asthma control. *Eur Respir J.* 1999;14:902-907. https://doi.org/10.1034/j.1399-3003.1999.14d29.x
- Juniper EF, Bousquet J, Abetz L, Bateman ED. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. *Respir Med.* 2006;100(4):616-621. https://doi.org/10.1016/j.rmed.2005.08.012
- Schmitt J, Langan S, Deckert S, et al. Assessment of clinical signs of atopic dermatitis: a systematic review and recommendation. *J Allergy Clin Immunol*. 2013;132(6):1337-1347. https://doi.org/10.1016/j.jaci.2013.07.008
- Simpson EL, Bieber T, Guttman-Yassky E, et al. Two Phase 3 trials of dupilumab versus placebo in atopic dermatitis. *N Engl J Med*. 2016;375(24):2335-2348. https://doi.org/10.1056/NEJMoa1610020
- Snaith RP. The Hospital Anxiety and Depression Scale. Health and Quality of Life Outcomes. 2003;1:29. Published August 01, 2003. Accessed July 29, 2022. http://www.hqlo.com/content/1/1/29

White D, Leach C, Sims R, et al. Validation of the Hospital Anxiety and Depression Scale for use with adolescents. *Br J Psychiatry*. 1999;175(5):452-454. https://doi.org/10.1192/bjp.175.5.452



Wright GJ, Cherwinski H, Foster-Cuevas M, et al. Characterization of the CD200 receptor family in mice and humans and their interactions with CD200. *J Immunol*. 2003;171(6):3034-3046. https://doi.org/10.4049/jimmunol.171.6.3034



Zigmond AS, Snaith RP. The Hospital Anxiety and Depression Scale. *Acta Psychiatr Scand*. 1983;67:361-370. https://doi.org/10.1111/j.1600-0447.1983.tb09716.x

# Signature Page for VV-CLIN-150737 v1.0

| Approval | PPD<br>PPD<br>06-May-2024 19:54:20 GMT+0000 |
|----------|---------------------------------------------|
| Approval | PPD<br>PPD<br>06-May-2024 19:57:40 GMT+0000 |

Signature Page for VV-CLIN-150737 v1.0